CLINICAL TRIAL: NCT01777295
Title: Development of Read-outs to Detect and Characterise the Early and Adaptive Immune Responses in Healthy, Hepatitis B Virus Naive Adults Vaccinated With the Hepatitis B Surface Antigen in Combination With a GSK Biologicals' Adjuvant System
Brief Title: Development of Read-outs in Healthy, Hepatitis B Virus Naive Adults Vaccinated With the Hepatitis B Surface Antigen (HBsAg) in Combination With a GlaxoSmithKline (GSK) Biologicals' Adjuvant System
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Collaborators: Region of Wallonia (Unknown); Public Private Partnership with Institute for Medical Immunology (Universite Libre de Bruxelles) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 116640; 2012-001344-22 (EudraCT Number)
Record Dates: First submitted 2013-01-24; First posted 2013-01-28 (Estimated); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-06

CONDITIONS: Hepatitis B
Keywords: Adults; Reactogenicity; Naive; Immune responses; Read-outs; Hepatitis B; Healthy
MeSH Terms: conditions — Hepatitis B | interventions — Hepatitis B Surface Antigens; Engerix-B

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBsAg/AS Group (Experimental): Subjects in this group received 1 dose of Placebo at Day -30 followed by 2 doses of HBsAg/AS, at Day 0 and Day 30.
  Interventions: Biological: Adjuvanted Hepatitis B surface antigen (HBsAg) candidate vaccine GSK2231392A.; Biological: Placebo
- Engerix-B Group (Active Comparator): Subjects in this group received 1 dose of Placebo at Day -30 followed by 3 doses of Engerix-B at Day 0, Day 30 and Day 180.
  Interventions: Biological: EngerixTM-B; Biological: Placebo

INTERVENTIONS:
Biological: Adjuvanted Hepatitis B surface antigen (HBsAg) candidate vaccine GSK2231392A. — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Other Names: HBsAg/AS
  Arms: HBsAg/AS Group
Biological: EngerixTM-B — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.
  Other Names: Engerix-B
  Arms: Engerix-B Group
Biological: Placebo — Intramuscular vaccination in the deltoid region of the non-dominant arm according to protocol schedule.

SUMMARY:
This study aims to develop innovative immunological read-outs and new technologies in order to further characterise the early immune response and its kinetics as well as the adaptive immune responses to adjuvanted vaccines.

This study will also evaluate the reactogenicity in healthy, hepatitis B virus naive adults vaccinated with the hepatitis B surface antigen in combination with a GSK Biologicals' Adjuvant System.

DETAILED DESCRIPTION:
This study will be conducted in 2 steps with 2 study groups in each step. The entire study period for Step 1 is from Day -30 to Day 210 (240 days) The entire study period for Step 2 is from Day 0 to Day 180 for Group C and from Day 0 to Day 330 for Group D.

Subjects will be blinded up to Day 60 in Step 1 and will be unblinded at the end of their Day 60 visit. Step 2 will be conducted in an open-label manner.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who, in the opinion of the investigator, can and will comply with the requirements of the protocol
* A male or female between, and including, 18 and 45 years of age at the time of first study product administration
* Written informed consent obtained from the subject
* Healthy subjects, in the opinion of the investigator, as established by medical history, clinical examination, and clinical laboratory assessment with no active disease that could interfere with the study endpoints, before entering into the study
* Body Mass Index (BMI) between 18.5 and 30 kg/m2
* Female subjects of non-childbearing potential may be enrolled in the study

  - Non-childbearing potential is defined as pre-menarche, current tubal ligation, hysterectomy, ovariectomy or post-menopause.
* Female subjects of childbearing potential may be enrolled in the study, if the subject:

  * has practiced adequate contraception for 30 days prior to first study product administration and
  * has a negative pregnancy test on the day of placebo administration/ vaccination, and
  * has agreed to continue adequate contraception during the entire treatment period and for 2 months after completion of the study.

Exclusion Criteria:

* Known history of HBV infection.
* Previous vaccination against hepatitis B.
* Positive for anti-hepatitis B surface (HBs) antibodies, anti-hepatitis B core (HBc) antibodies, HBsAg, HCV antibodies and/or HIV.
* Any previous administration of vaccine components.
* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccines within 30 days preceding the first study product administration, or planned use during the study period.
* No significant dietary restrictions or life-threatening food allergies.
* Regular use of non steroidal anti-inflammatory drugs within 1 month prior to first study product administration.
* Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs within 6 months prior to the first study product administration.. Inhaled and topical steroids are allowed.
* Planned administration / administration of a vaccine not foreseen by the study protocol in the period starting 30 days before the first study product administration and during the entire study period (both Steps), with the exception of the influenza vaccine (pandemic or seasonal) which can be administered > 21 days preceding or > 21 days following each placebo/vaccine administration.
* Administration of immunoglobulins and/or any blood products within the last 3 months preceding the first study product administration or planned administration during the study period.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including HIV based on screening evaluations and on medical history and physical examination.
* History of or current bleeding or coagulation disorder.
* Any known or clinical signs of anaemia or any clinical condition (including vascular disorder) that would preclude frequent blood drawings.
* Poor venous access as assessed at screening by the investigator.
* Blood loss, including blood donation, of more than 300 mL within 90 days before the first study product administration.
* History of or current autoimmune or other immune-mediated disease.
* Any haematological or biochemical level out of normal range before entering into the study, as follows:
* Haemoglobin level < lower normal limit (LNL).
* Platelet counts out of normal range.
* Alanine aminotransferase [ALT] > upper normal limit (UNL).
* Aspartate aminotransferase [AST] > UNL.
* Creatinine > UNL.
* c-reactive protein [CRP] > UNL.
* Creatine phosphokinase [CPK] > UNL without any plausible explanation for this abnormality (such as sport activity).

In case of haematological and/or biochemical value out of range for parameters mentioned here above, one re-testing of out of range value may be performed.

* Any acute or chronic, clinically significant disease, as determined by medical history, physical examination or laboratory screening tests.
* Known or suspected reaction or hypersensitivity likely to be exacerbated by any component of the vaccines.
* Acute disease and/or fever at the time of enrolment.
* Subjects with a minor illness (such as mild diarrhoea, mild upper respiratory infection) without fever may, be enrolled at the discretion of the investigator.
* Fever is defined as temperature ≥ 37.5°C for oral route.
* Pregnant or lactating female.
* Recent history of chronic alcohol consumption and/or drug abuse.
* Other conditions that the principal investigator judges may interfere with study findings.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2013-02-25 (Actual); Primary Completion 2016-05-17 (Actual); Study Completion 2016-09-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Antwerp, Belgium

REFERENCES:
- [Derived] Bechtold V, Smolen KK, Burny W, de Angelis SP, Delandre S, Essaghir A, Marchant A, Ndour C, Taton M, van der Most R, Willems F, Didierlaurent AM. Functional and epigenetic changes in monocytes from adults immunized with an AS01-adjuvanted vaccine. Sci Transl Med. 2024 Jul 31;16(758):eadl3381. doi: 10.1126/scitranslmed.adl3381. Epub 2024 Jul 31. PMID 39083587
- [Derived] Burny W, Herve C, Caubet M, Yarzabal JP, Didierlaurent AM. Utility of urinary cytokine levels as predictors of the immunogenicity and reactogenicity of AS01-adjuvanted hepatitis B vaccine in healthy adults. Vaccine. 2022 Apr 26;40(19):2714-2722. doi: 10.1016/j.vaccine.2022.03.050. Epub 2022 Mar 30. PMID 35367070
- [Derived] Burny W, Marchant A, Herve C, Callegaro A, Caubet M, Fissette L, Gheyle L, Legrand C, Ndour C, Tavares Da Silva F, van der Most R, Willems F, Didierlaurent AM, Yarzabal J; ECR-008 study group. Inflammatory parameters associated with systemic reactogenicity following vaccination with adjuvanted hepatitis B vaccines in humans. Vaccine. 2019 Mar 28;37(14):2004-2015. doi: 10.1016/j.vaccine.2019.02.015. Epub 2019 Mar 5. PMID 30850240

RESULTS

PARTICIPANT FLOW:
Groups:
- HBsAg/AS_1+2 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30, followed by 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30; or during Step 2 of the study, 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30. All vaccines were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
- Engerix-B_1+2 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30 followed by 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180; or during Step 2 of the study, 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180. All vaccine were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
Period: Overall Study
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Started | 40 | 41
Completed | 36 | 38
Not Completed | 4 | 3
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Pregnancy | 0 | 1
Not completed — Personal problem | 1 | 0
Not completed — Investigator call for AEs check | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- HBsAg/AS_1+2 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30, followed by 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30; and during Step 2 of the study, 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30. All vaccines were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
- Engerix-B_1+2 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30 followed by 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180; and during Step 2 of the study, 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180. All vaccine were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
- Total: Total of all reporting groups
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group | Total
Number analyzed (Participants) | 40 | 41 | 81
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.2 (4.1) | 37.5 (5.9) | 38.4 (5.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 26 | 51
  Male | 15 | 15 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Geographic ancestry: African Heritage / African American | 1 | 0 | 1
  Geographic ancestry: White - Arabic / North African Heritage | 1 | 2 | 3
  Geographic ancestry: White - Caucasian / European Heritage | 38 | 39 | 77

OUTCOME MEASURES:

1. Primary Outcome: Concentrations of Cytokines and Chemokines - Step 1
Description: Cytokines and chemokines analysed were E-selectin, granulocyte macrophage colony-stimulating factor (GM-CSF), interferon-γ (IFN-γ), interleukin-10 (IL-10), IL-18, IL-2, IL-3, IL-4, IL-5, IL-6, IL-6r, IL-7, IL-8, IFN-γ-inducible protein (IP-10), monocyte chemoattractant protein-1 (MCP-1), MCP-2, MCP-4, monokine induced by IFN-γ (MIG), macrophage inflammatory protein-1 alpha (MIP-1 alpha), MIP-1 beta, MIP3-alpha, MPIF-1, tumor necrosis factor-alpha (TNF-alpha) and TNF-beta. Concentrations are presented as median, expressed in picogram/milliliter (pg/mL), as measured by Multiplex in plasma.
Time Frame: At Day -30 prior to placebo administration
Population: Analyses were performed on the According-To-Protocol (ATP) cohort for innate immunogenicity up to Day 60 (step 1 only), which included all evaluable subjects, who complied with the protocol and for whom data concerning innate immunogenicity were available for at least one innate assay at one post-vaccination time point (up to Day 60).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- HBsAg/AS_1 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30, followed by 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30. All vaccines were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
- Engerix-B_1 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30 followed by 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180. All vaccine were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 6000 [4600 to 8300] | 6250 [4600 to 7800]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.5] | 3.3 [3.3 to 4.1]
  IL-18 | 198 [148 to 290] | 177 [152 to 215]
  IL-2 | 5.9 [5.9 to 7] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [20000 to 30000] | 22500 [22000 to 30000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.7 [4.2 to 6.6] | 5.1 [3.9 to 5.9]
  IP-10 | 225 [176 to 402] | 247.5 [195 to 280]
  MCP-1 | 107 [89 to 142] | 98.5 [83 to 117]
  MCP-2 | 18 [13 to 25] | 19.5 [17 to 26]
  MCP-4 | 1230 [1070 to 1550] | 1170 [1100 to 1600]
  MIG | 513 [354 to 682] | 435 [285 to 674]
  MIP-1 alpha | 20 [18 to 25] | 20 [18 to 24]
  MIP-1 beta | 190 [162 to 228] | 138 [126 to 205]
  MIP-3 alpha | 25 [11 to 32] | 18 [11 to 28]
  MPIF-1 | 1600 [1200 to 1800] | 1450 [1200 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

2. Primary Outcome: Cytokines and Chemokines Concentrations - Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 1.5 Hours
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5900 [4100 to 8500] | 6450 [4500 to 7600]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.7] | 3.3 [3.3 to 3.7]
  IL-18 | 172 [141 to 225] | 179.5 [136 to 215]
  IL-2 | 5.9 [5.9 to 7] | 5.9 [5.9 to 6.3]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [21000 to 30000] | 22000 [19000 to 29000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.2 [3.7 to 4.9] | 4.2 [3.2 to 5.3]
  IP-10 | 220 [183 to 330] | 207 [172 to 240]
  MCP-1 | 79 [58 to 101] | 77.5 [63 to 96]
  MCP-2 | 17 [13 to 24] | 19 [14 to 25]
  MCP-4 | 1300 [933 to 1480] | 1190 [896 to 1300]
  MIG | 392 [344 to 575] | 336 [269 to 487]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 19]
  MIP-1 beta | 141 [108 to 191] | 124.5 [107 to 151]
  MIP-3 alpha | 16 [13 to 27] | 16 [13 to 22]
  MPIF-1 | 1500 [1200 to 1600] | 1400 [1000 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

3. Primary Outcome: Concentrations of Cytokines and Chemokines in Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 3 Hours
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for innate immunogenicity up to Day 60 (step 1 only), which included all evaluable subjects, who complied with the protocol and for whom data concerning innate immunogenicity were available for at least one innate assay at one post-vaccination time point (up to Day 60).
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5600 [3800 to 7800] | 6300 [4100 to 7600]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.2] | 3.3 [3.3 to 3.4]
  IL-18 | 168 [154 to 283] | 173 [142 to 202]
  IL-2 | 5.9 [5.9 to 7.4] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 28000 [22000 to 34000] | 26000 [21000 to 33000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.2 [3.5 to 6.4] | 4 [3.2 to 5.3]
  IP-10 | 223 [169 to 396] | 217.5 [175 to 251]
  MCP-1 | 79 [65 to 92] | 64 [48 to 104]
  MCP-2 | 21 [14 to 27] | 20 [18 to 23]
  MCP-4 | 1170 [951 to 1440] | 1175 [1060 to 1310]
  MIG | 439 [347 to 558] | 343 [285 to 504]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 21]
  MIP-1 beta | 163 [120 to 199] | 127 [112 to 147]
  MIP-3 alpha | 18 [12 to 27] | 18 [14 to 22]
  MPIF-1 | 1600 [1200 to 1900] | 1300 [1000 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

4. Primary Outcome: Concentrations of Cytokines and Chemokines During Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 6 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5200 [3900 to 8300] | 6050 [4200 to 8100]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.6] | 3.3 [3.3 to 3.6]
  IL-18 | 176 [160 to 273] | 177.5 [132 to 233]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 2] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [21000 to 32000] | 24500 [20000 to 33000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.5 [3.7 to 6] | 4.5 [3.9 to 5.8]
  IP-10 | 217 [177 to 400] | 218 [174 to 252]
  MCP-1 | 104 [76 to 119] | 101 [76 to 129]
  MCP-2 | 18 [14 to 24] | 20.5 [16 to 23]
  MCP-4 | 1310 [1030 to 1570] | 1245 [1110 to 1490]
  MIG | 500 [320 to 614] | 378 [313 to 566]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 19]
  MIP-1 beta | 166 [140 to 215] | 146 [129 to 180]
  MIP-3 alpha | 21 [15 to 26] | 20 [15 to 24]
  MPIF-1 | 1500 [1200 to 1800] | 1400 [1100 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

5. Primary Outcome: Concentrations of Cytokines/Chemokines - Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 9 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5300 [3600 to 7100] | 6100 [4600 to 7500]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.8] | 3.3 [3.3 to 3.3]
  IL-18 | 173 [139 to 226] | 167.5 [117 to 202]
  IL-2 | 5.9 [5.9 to 14] | 5.9 [5.9 to 7.2]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 2.7] | 1.6 [1.6 to 1.6]
  IL-6r | 24000 [19000 to 31000] | 26000 [19000 to 29000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.9 [3.7 to 6.9] | 4.5 [3.6 to 5.3]
  IP-10 | 210 [162 to 327] | 205.5 [159 to 227]
  MCP-1 | 86 [65 to 104] | 81 [61 to 109]
  MCP-2 | 17 [15 to 24] | 17 [15 to 21]
  MCP-4 | 1310 [1050 to 1610] | 1145 [944 to 1400]
  MIG | 452 [313 to 610] | 327 [244 to 528]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 18]
  MIP-1 beta | 131 [111 to 185] | 119.5 [102 to 134]
  MIP-3 alpha | 19 [11 to 25] | 15 [11 to 17]
  MPIF-1 | 1400 [1100 to 1800] | 1200 [1000 to 1400]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

6. Primary Outcome: Concentrations of Cytokines/Chemokines in Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 12 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 5200 [3500 to 7900] | 5600 [4000 to 7800]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3] | 3.3 [3.3 to 3.3]
  IL-18 | 171 [150 to 244] | 180 [131 to 222]
  IL-2 | 5.9 [5.9 to 6.3] | 5.9 [5.9 to 6.3]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [21000 to 32000] | 24000 [21000 to 34000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.6 [3.9 to 5.9] | 4.5 [3.9 to 5.8]
  IP-10 | 217 [160 to 335] | 214 [182 to 246]
  MCP-1 | 117 [79 to 133] | 120 [96 to 137]
  MCP-2 | 18 [14 to 26] | 19 [17 to 25]
  MCP-4 | 1260 [1000 to 1480] | 1160 [997 to 1480]
  MIG | 460 [344 to 623] | 412 [341 to 564]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 21]
  MIP-1 beta | 159 [120 to 179] | 137 [118 to 167]
  MIP-3 alpha | 21 [14 to 26] | 22 [17 to 28]
  MPIF-1 | 1400 [1200 to 1700] | 1300 [1000 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

7. Primary Outcome: Concentrations of Cytokines/Chemokines During Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -30 plus 18 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 14 | 11
pg/mL
  E-selectin | 4950 [2900 to 6500] | 4200 [2700 to 6300]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.6] | 3.3 [3.3 to 3.3]
  IL-18 | 174 [118 to 267] | 142 [81 to 182]
  IL-2 | 6 [5.9 to 6.3] | 5.9 [5.9 to 6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 2.4]
  IL-6r | 21500 [18000 to 29000] | 21000 [18000 to 28000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.5 [4.6 to 8.2] | 6.1 [4.9 to 7.8]
  IP-10 | 243.5 [174 to 386] | 238 [170 to 483]
  MCP-1 | 98 [76 to 119] | 109 [79 to 132]
  MCP-2 | 18 [12 to 26] | 17 [16 to 27]
  MCP-4 | 1445 [1130 to 1640] | 1390 [1140 to 1710]
  MIG | 420 [373 to 636] | 458 [340 to 811]
  MIP-1 alpha | 18 [18 to 26] | 18 [18 to 23]
  MIP-1 beta | 143.5 [136 to 182] | 165 [128 to 216]
  MIP-3 alpha | 30 [21 to 34] | 20 [17 to 38]
  MPIF-1 | 1400 [1300 to 1700] | 1100 [920 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

8. Primary Outcome: Cytokines and Chemokines Concentrations in Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -29
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5900 [4300 to 8500] | 6350 [4500 to 8600]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.5] | 3.3 [3.3 to 3.3]
  IL-18 | 186 [149 to 261] | 177.5 [136 to 242]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.7] | 1.6 [1.6 to 1.7]
  IL-6r | 27000 [19000 to 35000] | 26500 [19000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.4 [3.9 to 6.9] | 5.2 [4.3 to 6.8]
  IP-10 | 241 [190 to 345] | 244.5 [200 to 307]
  MCP-1 | 93 [73 to 116] | 81.5 [66 to 104]
  MCP-2 | 19 [15 to 24] | 19 [16 to 25]
  MCP-4 | 1230 [1070 to 1350] | 1170 [1020 to 1450]
  MIG | 528 [327 to 695] | 418.5 [352 to 721]
  MIP-1 alpha | 19 [18 to 24] | 18 [18 to 21]
  MIP-1 beta | 169 [124 to 219] | 141.5 [123 to 188]
  MIP-3 alpha | 22 [17 to 28] | 21 [14 to 28]
  MPIF-1 | 1700 [1200 to 1900] | 1500 [1100 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

9. Primary Outcome: Cytokines and Chemokines Concetrations During Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -28
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5900 [3700 to 7800] | 6250 [4300 to 7900]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.9] | 3.3 [3.3 to 3.9]
  IL-18 | 182 [148 to 288] | 178.5 [120 to 232]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [20000 to 35000] | 25500 [20000 to 28000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.8 [3.7 to 6.5] | 4.9 [3.5 to 6.6]
  IP-10 | 270 [205 to 381] | 228 [186 to 304]
  MCP-1 | 74 [56 to 112] | 73.5 [47 to 90]
  MCP-2 | 19 [13 to 26] | 18.5 [15 to 26]
  MCP-4 | 1200 [937 to 1530] | 1140 [951 to 1340]
  MIG | 468 [336 to 568] | 397 [292 to 587]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 18]
  MIP-1 beta | 174 [141 to 227] | 151.5 [113 to 175]
  MIP-3 alpha | 20 [15 to 28] | 17.5 [11 to 33]
  MPIF-1 | 1500 [1200 to 1800] | 1350 [970 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

10. Primary Outcome: Cytokines/Chemokines Concentrations in Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -27
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 26 | 26
pg/mL
  E-selectin | 6150 [3700 to 8200] | 6250 [4000 to 7200]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.4 [3.3 to 4.5] | 3.3 [3.3 to 4.2]
  IL-18 | 183 [157 to 236] | 174.5 [139 to 217]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.7] | 1.6 [1.6 to 1.7]
  IL-6r | 26000 [21000 to 32000] | 24000 [21000 to 29000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.3 [3.4 to 6.6] | 4.2 [3.6 to 5.4]
  IP-10 | 239 [189 to 348] | 220.5 [186 to 281]
  MCP-1 | 84.5 [65 to 110] | 86.5 [73 to 109]
  MCP-2 | 18.5 [14 to 22] | 20 [15 to 25]
  MCP-4 | 1150 [989 to 1270] | 1060 [911 to 1360]
  MIG | 429.5 [349 to 542] | 403.5 [300 to 635]
  MIP-1 alpha | 18 [18 to 23] | 18 [18 to 19]
  MIP-1 beta | 165 [117 to 196] | 141 [106 to 181]
  MIP-3 alpha | 20.5 [18 to 27] | 21 [18 to 26]
  MPIF-1 | 1350 [1200 to 1700] | 1300 [1100 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

11. Primary Outcome: Cytokines and Chemokines Concentrations During Step 1
Description: as for outcome 1
Time Frame: Post-placebo at Day -23
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5500 [4000 to 8300] | 6150 [4700 to 7900]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.3] | 3.3 [3.3 to 3.5]
  IL-18 | 184 [150 to 247] | 176.5 [122 to 208]
  IL-2 | 5.9 [5.9 to 7] | 5.9 [5.9 to 7]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [17000 to 310000] | 23500 [19000 to 28000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.5 [3.9 to 6.8] | 5 [3.5 to 5.8]
  IP-10 | 241 [190 to 366] | 223 [186 to 285]
  MCP-1 | 88 [55 to 143] | 72 [66 to 96]
  MCP-2 | 15 [14 to 25] | 19 [16 to 23]
  MCP-4 | 1390 [1000 to 1480] | 1145 [1000 to 1350]
  MIG | 391 [337 to 524] | 375.5 [286 to 625]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 19]
  MIP-1 beta | 165 [128 to 199] | 138.5 [113 to 158]
  MIP-3 alpha | 21 [13 to 28] | 16 [10 to 21]
  MPIF-1 | 1600 [1200 to 1800] | 1350 [1000 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

12. Primary Outcome: Concentrations of Cytokines and Chemokines - Study Step 1
Description: as for outcome 1
Time Frame: Pre-dose1 at Day 0
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 6100 [4200 to 9000] | 6150 [5000 to 8600]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.5] | 3.3 [3.3 to 3.9]
  IL-18 | 169 [151 to 237] | 171 [119 to 207]
  IL-2 | 5.9 [5.9 to 6.5] | 5.9 [5.9 to 6.5]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [20000 to 32000] | 24500 [22000 to 29000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.9 [4.2 to 6.2] | 5 [4.2 to 7.4]
  IP-10 | 243 [199 to 294] | 225 [178 to 334]
  MCP-1 | 94 [75 to 121] | 92.5 [80 to 125]
  MCP-2 | 18 [14 to 22] | 19 [16 to 28]
  MCP-4 | 1310 [1110 to 1570] | 1260 [1030 to 1520]
  MIG | 496 [328 to 705] | 462.5 [303 to 701]
  MIP-1 alpha | 18 [18 to 23] | 18 [18 to 19]
  MIP-1 beta | 164 [121 to 198] | 153 [124 to 196]
  MIP-3 alpha | 20 [11 to 27] | 19.5 [14 to 24]
  MPIF-1 | 1500 [1300 to 1700] | 1300 [1000 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

13. Primary Outcome: Concentrations of Cytokines and Chemokines in Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 0 plus 1.5 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 5500 [4000 to 8400] | 5900 [4800 to 8100]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.8] | 3.3 [3.3 to 3.9]
  IL-18 | 168 [144 to 220] | 168 [126 to 208]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 7.4]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [21000 to 32000] | 25000 [19000 to 29000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.9 [3.6 to 5.5] | 4.2 [3.3 to 5.1]
  IP-10 | 224 [198 to 318] | 226 [186 to 265]
  MCP-1 | 74 [56 to 97] | 75 [56 to 108]
  MCP-2 | 18 [14 to 23] | 20 [16 to 22]
  MCP-4 | 1240 [943 to 1520] | 1240 [951 to 1340]
  MIG | 423 [385 to 535] | 378 [308 to 522]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 19]
  MIP-1 beta | 164 [132 to 194] | 137 [114 to 167]
  MIP-3 alpha | 18 [15 to 26] | 20 [14 to 24]
  MPIF-1 | 1500 [1300 to 1800] | 1200 [970 to 1400]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

14. Primary Outcome: Concentrations of Cytokines and Chemokines During Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 0 plus 6 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5400 [4100 to 7600] | 5900 [4300 to 7600]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3] | 3.3 [3.3 to 3.3]
  IL-18 | 170 [130 to 225] | 169 [110 to 220]
  IL-2 | 5.9 [5.9 to 6] | 5.9 [5.9 to 6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 3.4 [2.4 to 6] | 1.6 [1.6 to 1.7]
  IL-6r | 26000 [20000 to 33000] | 25000 [22000 to 30000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.6 [3.9 to 5.5] | 4.6 [3.9 to 7.2]
  IP-10 | 207 [179 to 270] | 204 [180 to 282]
  MCP-1 | 94 [75 to 123] | 85 [66 to 112]
  MCP-2 | 18 [15 to 20] | 18.5 [16 to 23]
  MCP-4 | 1130 [912 to 1390] | 1130 [989 to 1310]
  MIG | 459 [332 to 567] | 372.5 [302 to 557]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 19]
  MIP-1 beta | 165 [129 to 181] | 141 [111 to 174]
  MIP-3 alpha | 19 [15 to 28] | 18.5 [12 to 23]
  MPIF-1 | 1400 [1200 to 1600] | 1300 [1000 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

15. Primary Outcome: Cytokines and Chemokines Concentrations - Study Step 1
Description: as for outcome 1
Time Frame: Post-dose1 at Day 0 plus 12 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 5900 [4400 to 8800] | 6400 [5000 to 8000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.9 [3.3 to 5.5] | 3.3 [3.3 to 3.3]
  IL-18 | 171 [155 to 235] | 181.5 [128 to 205]
  IL-2 | 5.9 [5.9 to 6.5] | 5.9 [5.9 to 6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 6.3 [3.9 to 8.2] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [21000 to 32000] | 24000 [22000 to 33000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.2 [3.5 to 5.1] | 4.8 [4 to 5.6]
  IP-10 | 236 [197 to 281] | 194 [167 to 282]
  MCP-1 | 111 [87 to 137] | 111.5 [84 to 129]
  MCP-2 | 19 [15 to 27] | 19.5 [15 to 25]
  MCP-4 | 1260 [1000 to 1530] | 1265 [1030 to 1520]
  MIG | 478 [361 to 614] | 410 [296 to 588]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 19]
  MIP-1 beta | 183 [142 to 212] | 132 [102 to 171]
  MIP-3 alpha | 20 [17 to 28] | 19.5 [14 to 27]
  MPIF-1 | 1600 [1200 to 1700] | 1300 [1000 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

16. Primary Outcome: Cytokines and Chemokines Concentrations in Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 0 plus 18 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 14 | 11
pg/mL
  E-selectin | 5750 [3400 to 8000] | 4700 [3500 to 5900]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.8 [1.6 to 2.4] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.8] | 3.3 [3.3 to 3.3]
  IL-18 | 180 [155 to 217] | 126 [93 to 168]
  IL-2 | 5.9 [5.9 to 6] | 5.9 [5.9 to 6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 4.5 [3.1 to 6.9] | 1.6 [1.6 to 1.6]
  IL-6r | 22500 [17000 to 26000] | 22000 [19000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.9 [4.5 to 6.4] | 5.1 [4.2 to 6]
  IP-10 | 319 [268 to 477] | 228 [184 to 258]
  MCP-1 | 111 [91 to 130] | 115 [98 to 130]
  MCP-2 | 29.5 [19 to 34] | 20 [17 to 22]
  MCP-4 | 1400 [1310 to 1650] | 1400 [1220 to 1560]
  MIG | 571 [443 to 684] | 473 [367 to 722]
  MIP-1 alpha | 18 [18 to 20] | 18 [18 to 18]
  MIP-1 beta | 258 [200 to 303] | 134 [117 to 206]
  MIP-3 alpha | 35.5 [24 to 45] | 20 [17 to 30]
  MPIF-1 | 1850 [1500 to 2100] | 1400 [1100 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

17. Primary Outcome: Cytokines and Chemokines Concentrations During Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 1
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 26 | 25
pg/mL
  E-selectin | 5950 [4200 to 9500] | 6000 [4900 to 8900]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 5.2 [3.6 to 6.8] | 3.3 [3.3 to 3.6]
  IL-18 | 198.5 [167 to 267] | 181 [123 to 200]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 3 [1.6 to 4.1] | 1.6 [1.6 to 1.6]
  IL-6r | 26500 [22000 to 35000] | 24500 [21500 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.1 [4.1 to 6.3] | 4.4 [3.8 to 5.6]
  IP-10 | 295 [251 to 414] | 219 [179 to 326]
  MCP-1 | 85.5 [67 to 101] | 92 [73 to 112]
  MCP-2 | 21 [16 to 26] | 20 [17 to 25]
  MCP-4 | 1360 [1120 to 1600] | 1270 [1100 to 1630]
  MIG | 526 [441 to 678] | 425 [299 to 606]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 20]
  MIP-1 beta | 282.5 [234 to 408] | 145 [130 to 207]
  MIP-3 alpha | 17 [14 to 28] | 16 [12 to 23]
  MPIF-1 | 2300 [2000 to 2600] | 1400 [1200 to 1800]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

18. Primary Outcome: Cytokines/Chemokines Concentrations - Study Step 1
Description: as for outcome 1
Time Frame: Post-dose1 at Day 2
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 5800 [4300 to 9300] | 6300 [5000 to 7400]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.6 [3.3 to 4.3] | 3.3 [3.3 to 3.7]
  IL-18 | 219 [165 to 252] | 167 [130 to 219]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 25000 [18000 to 33000] | 24000 [20000 to 30000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.8 [3.8 to 6.4] | 5 [4.2 to 5.6]
  IP-10 | 455 [291 to 569] | 214 [174 to 303]
  MCP-1 | 83 [55 to 95] | 79 [58 to 101]
  MCP-2 | 22 [17 to 25] | 20 [15 to 25]
  MCP-4 | 1300 [1010 to 1600] | 1230 [1010 to 1390]
  MIG | 546 [435 to 593] | 364 [255 to 620]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 21]
  MIP-1 beta | 200 [160 to 265] | 149 [126 to 189]
  MIP-3 alpha | 19 [14 to 25] | 21 [16 to 28]
  MPIF-1 | 1600 [1300 to 2000] | 1300 [890 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

19. Primary Outcome: Cytokines/Chemokines Concentrations in Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 7
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 6600 [4100 to 8600] | 6700 [4800 to 8500]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.6 [3.3 to 4.9] | 3.3 [3.3 to 3.9]
  IL-18 | 202 [168 to 265] | 191 [126 to 231]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [21000 to 35000] | 25000 [21000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5 [4.2 to 6.9] | 5.1 [4.2 to 6.7]
  IP-10 | 235 [178 to 350] | 220.5 [185 to 279]
  MCP-1 | 94 [73 to 119] | 88.5 [71 to 125]
  MCP-2 | 20 [16 to 24] | 22.5 [18 to 30]
  MCP-4 | 1250 [1040 to 1390] | 1240 [1010 to 1420]
  MIG | 475 [384 to 582] | 436.5 [304 to 687]
  MIP-1 alpha | 18 [18 to 26] | 18 [18 to 22]
  MIP-1 beta | 171 [142 to 243] | 173.5 [146 to 213]
  MIP-3 alpha | 18 [14 to 26] | 22 [16 to 34]
  MPIF-1 | 1600 [1300 to 2100] | 1300 [1100 to 1500]
  TNF-alpha | 13 [13 to 17] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

20. Primary Outcome: Cytokines/Chemokines Concentrations During Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose1 at Day 30
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 6200 [4300 to 9000] | 6500 [5200 to 8000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.4] | 3.3 [3.3 to 3.4]
  IL-18 | 202 [151 to 248] | 183 [136 to 234]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 2.3] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [20000 to 32000] | 26000 [21000 to 30000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.8 [3.9 to 6] | 4.3 [3.4 to 5.8]
  IP-10 | 245 [211 to 349] | 235 [183 to 264]
  MCP-1 | 99 [72 to 136] | 86 [72 to 111]
  MCP-2 | 16 [14 to 23] | 20 [14 to 24]
  MCP-4 | 1180 [937 to 1340] | 1010 [937 to 1210]
  MIG | 475 [393 to 768] | 452 [281 to 691]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 18]
  MIP-1 beta | 175 [141 to 240] | 147 [126 to 181]
  MIP-3 alpha | 20 [15 to 30] | 20 [16 to 27]
  MPIF-1 | 1500 [1300 to 1800] | 1300 [940 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

21. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines - Step 1
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 1.5 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 6300 [3900 to 7600] | 5700 [4900 to 6800]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.5] | 3.3 [3.3 to 4.3]
  IL-18 | 171 [143 to 223] | 176 [127 to 207]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 24000 [18000 to 30000] | 25000 [20000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 3.2 [3 to 5.6] | 4.3 [2.7 to 5]
  IP-10 | 223 [189 to 336] | 215 [173 to 247]
  MCP-1 | 85 [58 to 112] | 87 [66 to 104]
  MCP-2 | 15 [12 to 23] | 18 [15 to 22]
  MCP-4 | 1250 [1030 to 1400] | 1090 [1020 to 1330]
  MIG | 421 [361 to 856] | 367 [269 to 575]
  MIP-1 alpha | 18 [18 to 22] | 18 [18 to 20]
  MIP-1 beta | 164 [132 to 196] | 136 [115 to 170]
  MIP-3 alpha | 17 [10 to 22] | 14 [11 to 19]
  MPIF-1 | 1400 [1200 to 1500] | 1200 [930 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

22. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines - Study Step 1
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 3 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 26 | 24
pg/mL
  E-selectin | 6550 [4000 to 8200] | 5700 [4450 to 6850]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 4.5] | 3.3 [3.3 to 3.4]
  IL-18 | 171.5 [146 to 204] | 158 [104 to 206.5]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 2.5] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [18000 to 31000] | 23000 [19000 to 28500]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.7 [3.9 to 6] | 4.5 [3.8 to 5]
  IP-10 | 208 [182 to 275] | 205.5 [176 to 243.5]
  MCP-1 | 75 [62 to 95] | 75 [51 to 85]
  MCP-2 | 15.5 [12 to 27] | 18 [14.5 to 22.5]
  MCP-4 | 1095 [979 to 1410] | 1085 [824.5 to 1250]
  MIG | 378.5 [313 to 513] | 358 [237 to 650.5]
  MIP-1 alpha | 18 [18 to 20] | 18 [18 to 18.5]
  MIP-1 beta | 153 [135 to 220] | 138 [123.5 to 157.5]
  MIP-3 alpha | 15 [10 to 22] | 14 [10 to 15.5]
  MPIF-1 | 1500 [1200 to 1600] | 1200 [980 to 1450]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

23. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines in Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 6 hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 26
pg/mL
  E-selectin | 6000 [4200 to 8100] | 5850 [4550 to 7000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.7] | 3.3 [3.3 to 3.3]
  IL-18 | 173.5 [151 to 227] | 183 [127.5 to 211.5]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 4.4 [2.8 to 6.7] | 1.6 [1.6 to 1.6]
  IL-6r | 23000 [18000 to 29000] | 24500 [20500 to 30500]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.2 [3.5 to 6.7] | 4.5 [3.5 to 5.2]
  IP-10 | 210.5 [182 to 248] | 196.5 [160 to 248.5]
  MCP-1 | 116.5 [98 to 132] | 95 [79 to 121]
  MCP-2 | 17 [12 to 24] | 18.5 [15 to 24]
  MCP-4 | 1245 [954 to 1590] | 1065 [936 to 1350]
  MIG | 375 [320 to 505] | 387.5 [239 to 671]
  MIP-1 alpha | 18 [18 to 19] | 18 [18 to 18]
  MIP-1 beta | 177.5 [128 to 225] | 139.5 [127.5 to 163.5]
  MIP-3 alpha | 16 [10 to 24] | 16 [12 to 22]
  MPIF-1 | 1400 [1200 to 1600] | 1300 [1015 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

24. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines During Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 9 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 24
pg/mL
  E-selectin | 6200 [4100 to 7400] | 5500 [4350 to 6850]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 5.2] | 3.3 [3.3 to 3.4]
  IL-18 | 177 [139 to 240] | 165 [115 to 229.5]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 6.6]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 4.8 [3.2 to 6.7] | 1.6 [1.6 to 1.6]
  IL-6r | 23000 [17000 to 30000] | 24500 [18500 to 30500]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.1 [3.2 to 5.5] | 4 [3.2 to 5.4]
  IP-10 | 217 [180 to 326] | 204 [168 to 234]
  MCP-1 | 103 [88 to 119] | 80 [55 to 106]
  MCP-2 | 18 [14 to 24] | 18.5 [14.5 to 20.5]
  MCP-4 | 1190 [999 to 1470] | 1075 [820 to 1295]
  MIG | 424 [384 to 621] | 350 [300 to 620]
  MIP-1 alpha | 18 [18 to 19] | 18 [18 to 18]
  MIP-1 beta | 167 [120 to 220] | 123.5 [108.5 to 146.5]
  MIP-3 alpha | 16 [14 to 23] | 15.5 [11 to 19]
  MPIF-1 | 1400 [1100 to 1600] | 1200 [950 to 1400]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

25. Primary Outcome: Plasma Concentrations of Cytokines/Chemokines During Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 12 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 25 | 25
pg/mL
  E-selectin | 5800 [4000 to 7800] | 5800 [4500 to 7000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 2.3 [1.6 to 3.1] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.8] | 3.3 [3.3 to 3.3]
  IL-18 | 166 [146 to 212] | 174 [124 to 220]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 6.4 [5 to 9] | 1.6 [1.6 to 1.7]
  IL-6r | 23000 [21000 to 31000] | 24000 [21000 to 32000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.9 [4.1 to 6] | 5.2 [3.2 to 6]
  IP-10 | 240 [228 to 335] | 200 [166 to 240]
  MCP-1 | 117 [96 to 150] | 95 [71 to 121]
  MCP-2 | 20 [14 to 26] | 18 [15 to 22]
  MCP-4 | 1100 [916 to 1330] | 1040 [852 to 1170]
  MIG | 499 [398 to 872] | 377 [290 to 689]
  MIP-1 alpha | 18 [18 to 20] | 18 [18 to 18]
  MIP-1 beta | 191 [162 to 238] | 134 [118 to 162]
  MIP-3 alpha | 20 [15 to 26] | 14 [11 to 20]
  MPIF-1 | 1500 [1100 to 1700] | 1300 [1100 to 1500]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

26. Primary Outcome: Plasma Concentrations of Cytokines/Chemokines - Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 30 plus 18 Hours
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 14 | 11
pg/mL
  E-selectin | 5400 [3400 to 8000] | 4500 [2900 to 5800]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 5.2 [1.6 to 7.4] | 1.6 [1.6 to 1.6]
  IL-10 | 4.5 [3.3 to 6] | 3.3 [3.3 to 3.4]
  IL-18 | 164.5 [151 to 241] | 168 [128 to 197]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 6.3 [4.2 to 8.3] | 1.6 [1.6 to 1.6]
  IL-6r | 19500 [13000 to 24000] | 24000 [17000 to 32000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 4.8 [4.1 to 5.4] | 5 [3.5 to 5.9]
  IP-10 | 589.5 [296 to 715] | 216 [196 to 430]
  MCP-1 | 104.5 [76 to 116] | 96 [91 to 106]
  MCP-2 | 33 [19 to 54] | 22 [16 to 23]
  MCP-4 | 1220 [1090 to 1290] | 1260 [1000 to 1340]
  MIG | 565.5 [373 to 791] | 442 [300 to 633]
  MIP-1 alpha | 18 [18 to 23] | 18 [18 to 23]
  MIP-1 beta | 283.5 [228 to 327] | 144 [111 to 176]
  MIP-3 alpha | 24 [19 to 31] | 17 [11 to 20]
  MPIF-1 | 1600 [1300 to 2300] | 1400 [1100 to 1700]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

27. Primary Outcome: Plasma Concentrations of Cytokines/Chemokines in Step 1 of Study
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 31
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 6800 [4300 to 8200] | 5800 [5200 to 7100]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 4.8 [1.7 to 8.6] | 1.6 [1.6 to 1.6]
  IL-10 | 4.8 [3.3 to 6.3] | 3.3 [3.3 to 3.3]
  IL-18 | 185 [151 to 258] | 166 [137 to 217]
  IL-2 | 8.5 [5.9 to 8.5] | 5.9 [5.9 to 8.5]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 3.6 [1.7 to 7.2] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [17000 to 33000] | 24000 [22000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.6 [4.8 to 7] | 4.8 [3.9 to 5.9]
  IP-10 | 763 [405 to 1130] | 212 [197 to 270]
  MCP-1 | 101 [79 to 137] | 71 [60 to 93]
  MCP-2 | 35 [19 to 67] | 17 [14 to 19]
  MCP-4 | 1250 [1090 to 1400] | 1090 [912 to 1330]
  MIG | 763 [604 to 1260] | 427 [308 to 597]
  MIP-1 alpha | 18 [18 to 21] | 18 [18 to 18]
  MIP-1 beta | 383 [301 to 540] | 142 [120 to 176]
  MIP-3 alpha | 22 [17 to 25] | 19 [12 to 28]
  MPIF-1 | 2000 [1500 to 2300] | 1100 [950 to 1600]
  TNF-alpha | 15 [13 to 21] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

28. Primary Outcome: Concentrations of Plasma Cytokines and Chemokines - Step 1
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 32
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 7000 [4400 to 9100] | 6000 [4900 to 8000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.5 [3.3 to 5.3] | 3.3 [3.3 to 3.5]
  IL-18 | 238 [195 to 269] | 190 [135 to 238]
  IL-2 | 5.9 [5.9 to 7] | 5.9 [5.9 to 7]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 2.5] | 1.6 [1.6 to 1.6]
  IL-6r | 27000 [21000 to 32000] | 24000 [21000 to 31000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.5 [4.3 to 6.5] | 5.1 [4 to 6.5]
  IP-10 | 760 [492 to 993] | 226 [192 to 276]
  MCP-1 | 75 [55 to 94] | 77 [65 to 121]
  MCP-2 | 24 [17 to 31] | 21 [17 to 25]
  MCP-4 | 1350 [1080 to 1580] | 1260 [1010 to 1560]
  MIG | 850 [667 to 1070] | 410 [320 to 581]
  MIP-1 alpha | 18 [18 to 19] | 18 [18 to 23]
  MIP-1 beta | 268 [222 to 307] | 142 [124 to 171]
  MIP-3 alpha | 23 [16 to 30] | 19 [13 to 28]
  MPIF-1 | 1800 [1400 to 2300] | 1200 [990 to 1700]
  TNF-alpha | 13 [13 to 14] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

29. Primary Outcome: Concentrations of Plasma Cytokines and Chemokines in Step 1
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 33
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 6400 [4400 to 8700] | 6300 [5100 to 8000]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.6] | 3.3 [3.3 to 3.6]
  IL-18 | 256 [195 to 351] | 181 [142 to 231]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 26000 [21000 to 33000] | 25000 [21000 to 28000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.5 [4.3 to 7.4] | 5.5 [4.3 to 6.2]
  IP-10 | 366 [288 to 524] | 249 [220 to 319]
  MCP-1 | 85 [65 to 101] | 93 [77 to 131]
  MCP-2 | 20 [16 to 28] | 20 [17 to 26]
  MCP-4 | 1390 [1190 to 1600] | 1280 [1090 to 1600]
  MIG | 796 [586 to 908] | 537 [456 to 722]
  MIP-1 alpha | 22 [18 to 24] | 19 [18 to 22]
  MIP-1 beta | 241 [175 to 279] | 163 [135 to 201]
  MIP-3 alpha | 25 [21 to 40] | 25 [21 to 32]
  MPIF-1 | 1800 [1400 to 2200] | 1300 [1100 to 1600]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3.4]

30. Primary Outcome: Concentrations of Plasma Cytokines and Chemokines During Step 1
Description: as for outcome 1
Time Frame: Post-dose 2 at Day 37
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
pg/mL
  E-selectin | 6200 [4000 to 8200] | 6000 [5000 to 7700]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3] | 3.3 [3.3 to 3.3]
  IL-18 | 194 [156 to 256] | 166 [123 to 196]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 28000 [16000 to 35000] | 25000 [20000 to 27000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.3 [3.9 to 6.6] | 5.5 [4.6 to 6]
  IP-10 | 259 [213 to 296] | 223 [179 to 289]
  MCP-1 | 83 [66 to 109] | 85 [63 to 99]
  MCP-2 | 17 [13 to 23] | 20 [16 to 24]
  MCP-4 | 1220 [1110 to 1480] | 1210 [1010 to 1340]
  MIG | 447 [398 to 535] | 364 [284 to 472]
  MIP-1 alpha | 18 [18 to 23] | 18 [18 to 19]
  MIP-1 beta | 150 [119 to 190] | 151 [126 to 175]
  MIP-3 alpha | 18 [15 to 28] | 18 [15 to 24]
  MPIF-1 | 1600 [1200 to 1800] | 1300 [1000 to 1400]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

31. Primary Outcome: Concentrations of Cytokines and Chemokines - Step 2
Description: as for outcome 1
Time Frame: Pre-dose 1 at Day 0
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for innate immunogenicity up to 30 days post last vaccination (step 2 only), which included all evaluable subjects, who complied with the protocol, and for whom data concerning innate immunogenicity were available for at least one innate assay at one post-vaccination time point.
Measure: Median (Inter-Quartile Range); unit: pg/mL
Groups:
- HBsAg/AS_2 Group: Subjects received, during Step 2 of the study, 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30. All vaccines were administered intramuscularly into the deltoid muscle of the non-dominant upper arm
- Engerix-B_2 Group: Subjects received, during Step 2 of the study, 3 doses of Engerix™-B vaccine at Day 0, Day 30 and Day 180. All vaccine were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 6 | 9
pg/mL
  E-selectin | 8100 [4200 to 8900] | 5400 [4400 to 5500]
  GM-CSF | 14 [14 to 14] | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.8] | 3.3 [3.3 to 3.3]
  IL-18 | 199.5 [175 to 377] | 179 [152 to 182]
  IL-2 | 5.9 [5.9 to 5.9] | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4] | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7] | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6] | 1.6 [1.6 to 1.6]
  IL-6r | 32000 [29000 to 36000] | 30000 [28000 to 36000]
  IL-7 | 8.2 [8.2 to 8.2] | 8.2 [8.2 to 8.2]
  IL-8 | 5.3 [3.5 to 11] | 4.4 [3.5 to 6.2]
  IP-10 | 300.5 [275 to 370] | 234 [166 to 278]
  MCP-1 | 86.5 [77 to 132] | 87 [67 to 96]
  MCP-2 | 22.5 [17 to 27] | 27 [19 to 30]
  MCP-4 | 1805 [1300 to 2010] | 2120 [1720 to 2260]
  MIG: number analyzed (Participants) | 0 | 0
  MIP-1 alpha | 18 [18 to 18] | 18 [18 to 18]
  MIP-1 beta | 234 [186 to 255] | 253 [200 to 300]
  MIP-3 alpha | 28.5 [23 to 64] | 29 [17 to 42]
  MPIF-1 | 1095 [820 to 1200] | 1100 [930 to 1200]
  TNF-alpha | 13 [13 to 13] | 13 [13 to 13]
  TNF-beta | 3 [3 to 3] | 3 [3 to 3]

32. Primary Outcome: Cytokines and Chemokines Concentrations - Step 2
Description: Cytokines and chemokines analysed were E-selectin, granulocyte macrophage colony-stimulating factor (GM-CSF), interferon-γ (IFN-γ), interleukin-10 (IL-10), IL-18, IL-2, IL-3, IL-4, IL-5, IL-6, IL-6r, IL-7, IL-8, IFN-γ-inducible protein (IP-10), monocyte chemoattractant protein-1 (MCP-1), MCP-2, MCP-4, monokine induced by IFN-γ (MIG), macrophage inflammatory protein-1 alpha (MIP-1 alpha), MIP-1 beta, MIP3-alpha, MPIF-1, tumor necrosis factor-alpha (TNF-alpha) and TNF-beta. Concentrations are presented as median, expressed in picogram/milliliter (pg/mL), as measured by Multiplex in plasma. The analysis was performed only on the HBsAg/AS_2 Group.
Time Frame: Post-dose 1 at Day 1
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_2 Group
Number analyzed (Participants) | 7
pg/mL
  E-selectin | 7900 [4300 to 9100]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.8 [3.3 to 4.7]
  IL-18 | 206 [182 to 260]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.7 [1.6 to 2.6]
  IL-6r | 24000 [22000 to 33000]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 3.9 [2.6 to 7.1]
  IP-10 | 294 [199 to 390]
  MCP-1 | 35 [27 to 114]
  MCP-2 | 26 [20 to 29]
  MCP-4 | 1240 [1130 to 1640]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 32]
  MIP-1 beta | 318 [241 to 391]
  MIP-3 alpha | 32 [17 to 46]
  MPIF-1 | 1400 [1200 to 1500]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

33. Primary Outcome: Concentrations of Cytokines and Chemokines During Step 2
Description: as for outcome 32
Time Frame: Post-dose 1 at Day 30
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_2 Group
Number analyzed (Participants) | 8
pg/mL
  E-selectin | 6200 [3600 to 8450]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.6]
  IL-18 | 166.5 [132.5 to 271.5]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 11.2]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.7]
  IL-6r | 29000 [24500 to 33500]
  IL-7 | 8.2 [8.2 to 10.1]
  IL-8 | 4.3 [3.1 to 8.4]
  IP-10 | 231.5 [160.5 to 318.5]
  MCP-1 | 46 [35 to 115.5]
  MCP-2 | 19.5 [17 to 20.5]
  MCP-4 | 1340 [1115 to 1450]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 172 [158.5 to 196.5]
  MIP-3 alpha | 25 [15 to 30.5]
  MPIF-1 | 1200 [855 to 1400]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

34. Primary Outcome: Concentrations of Cytokines and Chemokines in Step 2
Description: as for outcome 32
Time Frame: Post-dose2 at Day 30 plus 6 Hours
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_2 Group
Number analyzed (Participants) | 7
pg/mL
  E-selectin | 5400 [3400 to 8300]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3]
  IL-18 | 172 [150 to 247]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 10]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 3.7 [1.6 to 4.7]
  IL-6r | 34000 [27000 to 43000]
  IL-7 | 12 [8.2 to 21]
  IL-8 | 6.1 [3.6 to 9.1]
  IP-10 | 163 [128 to 205]
  MCP-1 | 59 [27 to 86]
  MCP-2 | 22 [18 to 25]
  MCP-4 | 1330 [979 to 1540]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 182 [154 to 266]
  MIP-3 alpha | 21 [13 to 28]
  MPIF-1 | 1300 [980 to 1700]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 6.3]

35. Primary Outcome: Concentrations of Cytokines/Chemokines - Step 2
Description: as for outcome 32
Time Frame: Post-dose 2 at Day 31
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_2 Group
Number analyzed (Participants) | 8
pg/mL
  E-selectin | 7450 [4600 to 10500]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 6.2 [3.4 to 17.6]
  IL-10 | 3.3 [3.3 to 4.4]
  IL-18 | 234 [181 to 339.5]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.7 [9.4 to 10]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 4 [2.2 to 5.7]
  IL-6r | 30500 [27000 to 41500]
  IL-7 | 10.1 [8.2 to 23.5]
  IL-8 | 7.9 [7.3 to 10.9]
  IP-10 | 737.5 [510 to 1270]
  MCP-1 | 142.5 [104 to 153]
  MCP-2 | 40.5 [32 to 72.5]
  MCP-4 | 1330 [974 to 1780]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 580 [359.5 to 780.5]
  MIP-3 alpha | 28 [19 to 39.5]
  MPIF-1 | 1750 [1500 to 1850]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

36. Primary Outcome: Concentrations of Cytokines/Chemokines in Step 2
Description: as for outcome 32
Time Frame: Post-dose 2 at Day 37
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | HBsAg/AS_2 Group
Number analyzed (Participants) | 8
pg/mL
  E-selectin | 6550 [3250 to 8450]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.8]
  IL-18 | 232 [145.5 to 322]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.7 [9.4 to 14]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.7]
  IL-6r | 28000 [26500 to 34500]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 8.5 [6.7 to 9.7]
  IP-10 | 170 [143 to 210]
  MCP-1 | 72.5 [27 to 104]
  MCP-2 | 18.5 [15 to 23]
  MCP-4 | 1275 [881.5 to 1635]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 174 [152.5 to 187.5]
  MIP-3 alpha | 17 [11.5 to 94]
  MPIF-1 | 1100 [995 to 1450]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 11.2]

37. Primary Outcome: Concentrations of Cytokines/Chemokines During Step 2
Description: Cytokines and chemokines analysed were E-selectin, granulocyte macrophage colony-stimulating factor (GM-CSF), interferon-γ (IFN-γ), interleukin-10 (IL-10), IL-18, IL-2, IL-3, IL-4, IL-5, IL-6, IL-6r, IL-7, IL-8, IFN-γ-inducible protein (IP-10), monocyte chemoattractant protein-1 (MCP-1), MCP-2, MCP-4, monokine induced by IFN-γ (MIG), macrophage inflammatory protein-1 alpha (MIP-1 alpha), MIP-1 beta, MIP3-alpha, MPIF-1, tumor necrosis factor-alpha (TNF-alpha) and TNF-beta. Concentrations are presented as median, expressed in picogram/milliliter (pg/mL), as measured by Multiplex in plasma.
  The analysis was performed only on the Engerix-B_2 Group.
Time Frame: Post-dose 2 at Day 180
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Engerix-B_2 Group
Number analyzed (Participants) | 9
pg/mL
  E-selectin | 4900 [4300 to 5800]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3]
  IL-18 | 159 [144 to 190]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6]
  IL-6r | 24000 [24000 to 32000]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 4.4 [3.5 to 5.3]
  IP-10 | 156 [121 to 260]
  MCP-1 | 77 [57 to 77]
  MCP-2 | 20 [14 to 27]
  MCP-4 | 1640 [1540 to 1810]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 189 [177 to 257]
  MIP-3 alpha | 25 [13 to 32]
  MPIF-1 | 920 [830 to 970]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

38. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines - Study Step 2
Description: Cytokines and chemokines analysed were E-selectin, granulocyte macrophage colony-stimulating factor (GM-CSF), interferon-γ (IFN-γ), interleukin-10 (IL-10), IL-18, IL-2, IL-3, IL-4, IL-5, IL-6, IL-6r, IL-7, IL-8, IFN-γ-inducible protein (IP-10), monocyte chemoattractant protein-1 (MCP-1), MCP-2, MCP-4, monokine induced by IFN-γ (MIG), macrophage inflammatory protein-1 alpha (MIP-1 alpha), MIP-1 beta, MIP3-alpha, MPIF-1, tumor necrosis factor-alpha (TNF-alpha) and TNF-beta. Concentrations are presented as median, expressed in picogram/milliliter (pg/mL), as measured by Multiplex in plasma.The analysis was performed only on theEngerix-B_2 Group.
Time Frame: Post-dose 3 at Day 180 plus 6 Hours
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Engerix-B_2 Group
Number analyzed (Participants) | 9
pg/mL
  E-selectin | 4600 [4100 to 5800]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3]
  IL-18 | 144 [133 to 152]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6]
  IL-6r | 25000 [24000 to 30000]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 3.5 [2.6 to 4.4]
  IP-10 | 145 [105 to 214]
  MCP-1 | 46 [35 to 67]
  MCP-2 | 22 [15 to 26]
  MCP-4 | 1640 [1350 to 1720]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 193 [175 to 211]
  MIP-3 alpha | 21 [15 to 25]
  MPIF-1 | 890 [840 to 1100]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

39. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines in Step 2 of Study
Description: as for outcome 37
Time Frame: Post-dose 3 at Day 181
Population: as for outcome 31
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Engerix-B_2 Group
Number analyzed (Participants) | 8
pg/mL
  E-selectin | 4900 [4300 to 5900]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.8]
  IL-18 | 152 [140.5 to 192]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 11.2]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6]
  IL-6r | 24500 [22500 to 31500]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 3.5 [2.6 to 3.5]
  IP-10 | 152 [119.5 to 211.5]
  MCP-1 | 67 [35 to 86.5]
  MCP-2 | 19.5 [13 to 25.5]
  MCP-4 | 1720 [1390 to 1790]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 173.5 [166.5 to 213]
  MIP-3 alpha | 17 [15 to 21]
  MPIF-1 | 875 [745 to 1100]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

40. Primary Outcome: Plasma Concentrations of Cytokines and Chemokines During Step 2 of Study
Description: as for outcome 37
Time Frame: Post-dose 3 at Day 187
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: pg/mL
Arm/Group | Engerix-B_2 Group
Number analyzed (Participants) | 5
pg/mL
  E-selectin | 4600 [4200 to 5500]
  GM-CSF | 14 [14 to 14]
  IFN-γ | 1.6 [1.6 to 1.6]
  IL-10 | 3.3 [3.3 to 3.3]
  IL-18 | 163 [137 to 167]
  IL-2 | 5.9 [5.9 to 5.9]
  IL-3 | 1.6 [1.6 to 1.6]
  IL-4 | 9.4 [9.4 to 9.4]
  IL-5 | 2.7 [2.7 to 2.7]
  IL-6 | 1.6 [1.6 to 1.6]
  IL-6r | 30000 [26000 to 35000]
  IL-7 | 8.2 [8.2 to 8.2]
  IL-8 | 3.5 [3.5 to 4.4]
  IP-10 | 201 [107 to 201]
  MCP-1 | 35 [35 to 35]
  MCP-2 | 22 [17 to 25]
  MCP-4 | 1810 [1720 to 2120]
  MIG: number analyzed (Participants) | 0
  MIP-1 alpha | 18 [18 to 18]
  MIP-1 beta | 175 [175 to 193]
  MIP-3 alpha | 17 [17 to 25]
  MPIF-1 | 820 [750 to 970]
  TNF-alpha | 13 [13 to 13]
  TNF-beta | 3 [3 to 3]

41. Secondary Outcome: Anti-Hepatitis B Surface (Anti-HBs) Antibody Concentrations in Serum - Step 1
Description: Anti-HBs antibody concentrations in serum were measured by Chemi Luminiscence Immuno Assay (CLIA). Concentrations were presented as geometric mean concentrations, in milli-International Units per milliliter (mIU/mL).
Time Frame: At Day 0 (PRE) and Day 60 (D60) post-vaccination
Population: The analysis was performed on the ATP cohort for adaptive immunogenicity up to Day 60 (step 1 only) which included all evaluable subjects who complied with the protocol and for whom data concerning adaptive immunogenicity were available for at least one adaptive assay at one post-vaccination time point (up to Day 60).
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 25
mIU/mL
  Anti-HBs, PRE (D0) | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Anti-HBs, PII (D60) | 3322.4 [2332.2 to 4733.0] | 35.8 [11.6 to 111.1]

42. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Step 1
Description: Assessed solicited local symptoms were pain, redness and swelling. Any = occurrence of the symptom regardless of intensity grade. Grade 3 pain = pain that prevented normal activity. Grade 3 redness/swelling = redness/swelling spreading beyond 100 millimeters (mm) of injection site.
Time Frame: During the 7-day (Days 0-6) post-placebo (PP) and post-vaccination period following each vaccine dose (D1 and D2) and across doses
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented, who have filled in their symptom sheets.
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  Any pain, PP | 2 | 3
  Grade 3 pain, PP | 0 | 1
  Any redness, PP | 0 | 0
  Grade 3 redness, PP | 0 | 0
  Any swelling, PP | 0 | 0
  Grade 3 swelling, PP | 0 | 0
  Any pain, D1: number analyzed (Participants) | 28 | 28
  Any pain, D1 | 18 | 7
  Grade 3 pain, D1: number analyzed (Participants) | 28 | 28
  Grade 3 pain, D1 | 0 | 0
  Any redness, D1: number analyzed (Participants) | 28 | 28
  Any redness, D1 | 6 | 1
  Grade 3 redness, D1: number analyzed (Participants) | 28 | 28
  Grade 3 redness, D1 | 0 | 0
  Any swelling, D1: number analyzed (Participants) | 28 | 28
  Any swelling, D1 | 4 | 0
  Grade 3 swelling, D1: number analyzed (Participants) | 28 | 28
  Grade 3 swelling, D1 | 0 | 0
  Any pain, D2: number analyzed (Participants) | 27 | 28
  Any pain, D2 | 15 | 6
  Grade 3 pain, D2: number analyzed (Participants) | 27 | 28
  Grade 3 pain, D2 | 0 | 1
  Any redness, D2: number analyzed (Participants) | 27 | 28
  Any redness, D2 | 5 | 0
  Grade 3 redness, D2: number analyzed (Participants) | 27 | 28
  Grade 3 redness, D2 | 1 | 0
  Any swelling, D2: number analyzed (Participants) | 27 | 28
  Any swelling, D2 | 1 | 0
  Grade 3 swelling, D2: number analyzed (Participants) | 27 | 28
  Grade 3 swelling, D2 | 0 | 0
  Any pain, Across Doses: number analyzed (Participants) | 28 | 28
  Any pain, Across Doses | 21 | 8
  Grade 3 pain, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 pain, Across Doses | 0 | 1
  Any redness, Across Doses: number analyzed (Participants) | 28 | 28
  Any redness, Across Doses | 8 | 1
  Grade 3 redness, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 redness, Across Doses | 1 | 0
  Any swelling, Across Doses: number analyzed (Participants) | 28 | 28
  Any swelling, Across Doses | 4 | 0
  Grade 3 swelling, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 swelling, Across Doses | 0 | 0

43. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms - Step 1
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms [nausea, vomiting, diarrhoea and /or abdominal pain], headache, malaise, myalgia, shivering and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination
Time Frame: as for outcome 42
Population: as for outcome 42
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  Any fatigue, PP | 8 | 12
  Grade 3 fatigue, PP | 0 | 1
  Related fatigue, PP | 2 | 2
  Any gastrointestinal symptoms, PP | 8 | 8
  Grade 3 gastrointestinal symptoms, PP | 0 | 2
  Related gastrointestinal symptoms, PP | 1 | 0
  Any headache, PP | 11 | 13
  Grade 3 headache, PP | 0 | 1
  Related headache, PP | 2 | 2
  Any malaise, PP | 3 | 4
  Grade 3 malaise, PP | 0 | 0
  Related malaise, PP | 0 | 1
  Any myalgia, PP | 2 | 5
  Grade 3 myalgia, PP | 0 | 1
  Related myalgia, PP | 1 | 0
  Any shivering, PP | 4 | 3
  Grade 3 shivering, PP | 0 | 1
  Related shivering, PP | 0 | 0
  Any temperature, PP | 1 | 2
  Grade 3 temperature, PP | 0 | 0
  Related temperature, PP | 0 | 0
  Any Fatigue, D1: number analyzed (Participants) | 28 | 28
  Any Fatigue, D1 | 3 | 6
  Grade 3 fatigue, D1: number analyzed (Participants) | 28 | 28
  Grade 3 fatigue, D1 | 1 | 0
  Related fatigue, D1: number analyzed (Participants) | 28 | 28
  Related fatigue, D1 | 2 | 6
  Any gastrointestinal symptoms, D1: number analyzed (Participants) | 28 | 28
  Any gastrointestinal symptoms, D1 | 4 | 6
  Grade 3 gastrointestinal symptoms, D1: number analyzed (Participants) | 28 | 28
  Grade 3 gastrointestinal symptoms, D1 | 0 | 1
  Related gastrointestinal symptoms, D1: number analyzed (Participants) | 28 | 28
  Related gastrointestinal symptoms, D1 | 4 | 3
  Any headache, D1: number analyzed (Participants) | 28 | 28
  Any headache, D1 | 14 | 5
  Grade 3 headache, D1: number analyzed (Participants) | 28 | 28
  Grade 3 headache, D1 | 0 | 1
  Related headache, D1: number analyzed (Participants) | 28 | 28
  Related headache, D1 | 11 | 4
  Any malaise, D1: number analyzed (Participants) | 28 | 28
  Any malaise, D1 | 4 | 2
  Grade 3 malaise, D1: number analyzed (Participants) | 28 | 28
  Grade 3 malaise, D1 | 0 | 0
  Related malaise, D1: number analyzed (Participants) | 28 | 28
  Related malaise, D1 | 4 | 2
  Any myalgia, D1: number analyzed (Participants) | 28 | 28
  Any myalgia, D1 | 10 | 1
  Grade 3 myalgia, D1: number analyzed (Participants) | 28 | 28
  Grade 3 myalgia, D1 | 0 | 0
  Related myalgia, D1: number analyzed (Participants) | 28 | 28
  Related myalgia, D1 | 9 | 1
  Any shivering, D1: number analyzed (Participants) | 28 | 28
  Any shivering, D1 | 2 | 0
  Grade 3 shivering, D1: number analyzed (Participants) | 28 | 28
  Grade 3 shivering, D1 | 0 | 0
  Related shivering, D1: number analyzed (Participants) | 28 | 28
  Related shivering, D1 | 2 | 0
  Any temperature (≥37.5 °C), D1: number analyzed (Participants) | 28 | 28
  Any temperature (≥37.5 °C), D1 | 2 | 1
  Grade 3 temperature (> 39.5 °C), D1: number analyzed (Participants) | 28 | 28
  Grade 3 temperature (> 39.5 °C), D1 | 0 | 0
  Related temperature, D1: number analyzed (Participants) | 28 | 28
  Related temperature, D1 | 1 | 0
  Any Fatigue, D2: number analyzed (Participants) | 27 | 28
  Any Fatigue, D2 | 10 | 8
  Grade 3 fatigue, D2: number analyzed (Participants) | 27 | 28
  Grade 3 fatigue, D2 | 1 | 0
  Related fatigue, D2: number analyzed (Participants) | 27 | 28
  Related fatigue, D2 | 10 | 7
  Any gastrointestinal symptoms, D2: number analyzed (Participants) | 27 | 28
  Any gastrointestinal symptoms, D2 | 4 | 5
  Grade 3 gastrointestinal symptoms, D2: number analyzed (Participants) | 27 | 28
  Grade 3 gastrointestinal symptoms, D2 | 0 | 3
  Related gastrointestinal symptoms, D2: number analyzed (Participants) | 27 | 28
  Related gastrointestinal symptoms, D2 | 4 | 5
  Any headache, D2: number analyzed (Participants) | 27 | 28
  Any headache, D2 | 14 | 5
  Grade 3 headache, D2: number analyzed (Participants) | 27 | 28
  Grade 3 headache, D2 | 0 | 1
  Related headache, D2: number analyzed (Participants) | 27 | 28
  Related headache, D2 | 14 | 5
  Any malaise, D2: number analyzed (Participants) | 27 | 28
  Any malaise, D2 | 7 | 6
  Grade 3 malaise, D2: number analyzed (Participants) | 27 | 28
  Grade 3 malaise, D2 | 2 | 1
  Related malaise, D2: number analyzed (Participants) | 27 | 28
  Related malaise, D2 | 7 | 6
  Any myalgia, D2: number analyzed (Participants) | 27 | 28
  Any myalgia, D2 | 10 | 2
  Grade 3 myalgia, D2: number analyzed (Participants) | 27 | 28
  Grade 3 myalgia, D2 | 0 | 0
  Related myalgia, D2: number analyzed (Participants) | 27 | 28
  Related myalgia, D2 | 10 | 1
  Any shivering, D2: number analyzed (Participants) | 27 | 28
  Any shivering, D2 | 9 | 2
  Grade 3 shivering, D2: number analyzed (Participants) | 27 | 28
  Grade 3 shivering, D2 | 0 | 0
  Related shivering, D2: number analyzed (Participants) | 27 | 28
  Related shivering, D2 | 9 | 2
  Any temperature (≥37.5 °C), D2: number analyzed (Participants) | 27 | 28
  Any temperature (≥37.5 °C), D2 | 5 | 1
  Grade 3 temperature (> 39.5 °C), D2: number analyzed (Participants) | 27 | 28
  Grade 3 temperature (> 39.5 °C), D2 | 0 | 0
  Related temperature, D2: number analyzed (Participants) | 27 | 28
  Related temperature, D2 | 4 | 0
  Any Fatigue, Across Doses: number analyzed (Participants) | 28 | 28
  Any Fatigue, Across Doses | 10 | 9
  Grade 3 fatigue, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 fatigue, Across Doses | 2 | 0
  Related fatigue, Across Doses: number analyzed (Participants) | 28 | 28
  Related fatigue, Across Doses | 10 | 9
  Any gastrointestinal symptoms, Across Doses: number analyzed (Participants) | 28 | 28
  Any gastrointestinal symptoms, Across Doses | 8 | 8
  Grade 3 gastrointestinal symptoms, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 gastrointestinal symptoms, Across Doses | 0 | 4
  Related gastrointestinal symptoms, Across Doses: number analyzed (Participants) | 28 | 28
  Related gastrointestinal symptoms, Across Doses | 8 | 7
  Any headache, Across Doses: number analyzed (Participants) | 28 | 28
  Any headache, Across Doses | 17 | 6
  Grade 3 headache, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 headache, Across Doses | 0 | 1
  Related headache, Across Doses: number analyzed (Participants) | 28 | 28
  Related headache, Across Doses | 15 | 6
  Any malaise, Across Doses: number analyzed (Participants) | 28 | 28
  Any malaise, Across Doses | 8 | 7
  Grade 3 malaise, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 malaise, Across Doses | 2 | 1
  Related malaise, Across Doses: number analyzed (Participants) | 28 | 28
  Related malaise, Across Doses | 8 | 7
  Any myalgia, Across Doses: number analyzed (Participants) | 28 | 28
  Any myalgia, Across Doses | 14 | 2
  Grade 3 myalgia, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 myalgia, Across Doses | 0 | 0
  Related myalgia, Across Doses: number analyzed (Participants) | 28 | 28
  Related myalgia, Across Doses | 13 | 2
  Any shivering, Across Doses: number analyzed (Participants) | 28 | 28
  Any shivering, Across Doses | 10 | 2
  Grade 3 shivering, Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 shivering, Across Doses | 0 | 0
  Related shivering, Across Doses: number analyzed (Participants) | 28 | 28
  Related shivering, Across Doses | 10 | 2
  Any temperature (≥37.5 °C), Across Doses: number analyzed (Participants) | 28 | 28
  Any temperature (≥37.5 °C), Across Doses | 6 | 2
  Grade 3 temperature (> 39.5 °C), Across Doses: number analyzed (Participants) | 28 | 28
  Grade 3 temperature (> 39.5 °C), Across Doses | 0 | 0
  Related temperature, Across Doses: number analyzed (Participants) | 28 | 28
  Related temperature, Across Doses | 4 | 0

44. Secondary Outcome: Number of Subjects With Solicited Symptoms, as Assessed by the Investigator/Study Nurse - Step 1
Description: Assessed solicited symptoms were fever [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)], pain, redness [spreading beyond 20 millimeters (mm) of injection site], induration [spreading beyond 20 millimeters (mm) of injection site], swelling [spreading beyond 20 millimeters (mm) of injection site] and muscle stiffness.
Time Frame: Up to 4 days post-placebo/vaccine administration.
Population: The analysis was performed on the Total Vaccinated cohort, which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  Fever (≥37.5), placebo | 0 | 0
  Fever (≥37.5), D1: number analyzed (Participants) | 28 | 30
  Fever (≥37.5), D1 | 2 | 2
  Fever (≥37.5), D2: number analyzed (Participants) | 27 | 28
  Fever (≥37.5), D2 | 8 | 0
  Pain, placebo | 1 | 4
  Pain, D1: number analyzed (Participants) | 28 | 30
  Pain, D1 | 19 | 9
  Pain, D2: number analyzed (Participants) | 27 | 28
  Pain, D2 | 19 | 8
  Redness, placebo | 0 | 0
  Redness, D1: number analyzed (Participants) | 28 | 30
  Redness, D1 | 8 | 1
  Redness, D2: number analyzed (Participants) | 27 | 28
  Redness, D2 | 7 | 0
  Induration, placebo | 0 | 0
  Induration, D1: number analyzed (Participants) | 28 | 30
  Induration, D1 | 0 | 0
  Induration, D2: number analyzed (Participants) | 27 | 28
  Induration, D2 | 1 | 0
  Swelling, placebo | 0 | 0
  Swelling, D1: number analyzed (Participants) | 28 | 30
  Swelling, D1 | 3 | 1
  Swelling, D2: number analyzed (Participants) | 27 | 28
  Swelling, D2 | 4 | 1
  Muscle stiffness, placebo | 0 | 2
  Muscle stiffness, D1: number analyzed (Participants) | 28 | 30
  Muscle stiffness, D1 | 14 | 5
  Muscle stiffness, D2: number analyzed (Participants) | 27 | 28
  Muscle stiffness, D2 | 15 | 4

45. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Step 1
Description: An unsolicited AE covers any untoward medical occurrence in a clinical investigation subject temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset out-side the specified period of follow-up for solicited symptoms. Any was defined as the occurrence of any unsolicited AE regardless of intensity grade or relation to vaccination.
Time Frame: Within the 28-day (Days 0-27) post-placebo (PP) and post-product administration period.
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  Any AEs, post-placebo | 12 | 16
  Any AEs, post-product administration: number analyzed (Participants) | 28 | 29
  Any AEs, post-product administration | 14 | 15

46. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Step 1
Description: Serious adverse events (SAEs) assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization or result in disability/incapacity.
Time Frame: From Day 0 up to Day 60 for the HBsAg/AS_1 Group and from Day 0 up to Day 210 for the Engerix-B_1 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  Day 60 SAEs | 0 | 0
  Day 210 SAEs: number analyzed (Participants) | 0 | 30
  Day 210 SAEs | 0 | 1

47. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Disorders (pIMDs) - Step 1
Description: PIMD(s) are a subset of AEs that include autoimmune diseases and other inflammatory and/or neurologic disorders of interest which may or may not have an autoimmune aetiology.
Time Frame: From Day 0 up to Day 60 for the HBsAg/AS_1 Group and from Day 0 up to Day 210 for the Engerix-B_1 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  pIMDs - Day 60 | 0 | 0
  pIMDs - Day 210: number analyzed (Participants) | 0 | 30
  pIMDs - Day 210 | 0 | 0

48. Secondary Outcome: Number of Subjects With Any New Medical Conditions Requiring Medical Attention (MAEs) - Step 1
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination. Analysis of intensity and relationship to vaccination of MAEs was not performed.
Time Frame: From Day 0 up to Day 60 for the HBsAg/AS_1 Group and from Day 0 up to Day 210 for the Engerix-B_1 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
Participants
  MAEs - Day 60 | 0 | 0
  MAEs - Day 210: number analyzed (Participants) | 0 | 30
  MAEs - Day 210 | 0 | 1

49. Secondary Outcome: Levels of Alanine Aminotransferase (ALT) in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included ALT levels. ALT concentrations were expressed in units per liter (U/L). ALT levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: At Day 0, Day 0 H6, Day 0 H12, Day 0 H18, Day 1, Day 7, Day 30, Day 30 H6, Day 30 H12, Day 30 H18, Day 31, Day 37 and Day 60
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
U/L
  ALT, Dose 1, Day 0 | 27.5 [22.5 to 32.5] | 27 [23 to 31]
  ALT, Dose 1 (Day 0 H6) | 26.5 [22 to 33] | 26 [22 to 34]
  ALT, Dose 1 (Day 0 H12) | 27 [23.5 to 31.5] | 26 [24 to 33]
  ALT, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  ALT, Dose 1 (Day 0 H18) | 28 [25 to 35] | 24 [16 to 48]
  ALT, Dose 1, Day 1 | 25.5 [20 to 33] | 27 [20 to 35]
  ALT, Dose 1, Day 7 | 26.5 [22 to 32.5] | 28 [19 to 34]
  ALT, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  ALT, Dose 2, Day 30 | 27 [22 to 36] | 30 [24 to 33]
  ALT, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  ALT, Dose 2 (Day 30 H6) | 27 [23 to 34] | 28 [25 to 32]
  ALT, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  ALT, Dose 2 (Day 30 H12) | 27 [24 to 34] | 28 [23 to 33.5]
  ALT, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  ALT, Dose 2 (Day 30 H18) | 32 [25 to 37] | 26 [24 to 46]
  ALT, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  ALT, Dose 2, Day 31 | 27 [22 to 33] | 27 [23 to 34]
  ALT, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  ALT, Dose 2, Day 37 | 27 [22 to 30] | 26 [23.5 to 33]
  ALT, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  ALT, Dose 2, Day 60 | 28 [23 to 32] | 28 [22.5 to 36]

50. Secondary Outcome: Levels of Aspartate Aminotransferase (AST) in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included AST levels. AST concentrations were expressed in units per liter (U/L). AST levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
U/L
  AST, Dose 1, Day 0 | 21 [18 to 26] | 23 [18 to 25]
  AST, Dose 1 (Day 0 H6) | 20.5 [18.5 to 24] | 21 [17 to 25]
  AST, Dose 1 (Day 0 H12) | 20 [18.5 to 22.5] | 20 [17 to 25]
  AST, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  AST, Dose 1 (Day 0 H18) | 19 [15 to 24] | 18 [17 to 28]
  AST, Dose 1, Day 1 | 19 [16 to 22.5] | 20 [18 to 23]
  AST, Dose 1, Day 7 | 21 [18.5 to 25.5] | 21 [18 to 29]
  AST, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  AST, Dose 2, Day 30 | 21 [19 to 26] | 23 [19 to 25]
  AST, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 29
  AST, Dose 2 (Day 30 H6) | 21 [19 to 24] | 22 [20 to 25.5]
  AST, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 29
  AST, Dose 2 (Day 30 H12) | 20 [18 to 25] | 21 [20 to 24.5]
  AST, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  AST, Dose 2 (Day 30 H18) | 20 [19 to 22] | 19.5 [16 to 30]
  AST, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  AST, Dose 2, Day 31 | 19 [17 to 23] | 21 [18 to 25.5]
  AST, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  AST, Dose 2, Day 37 | 22 [19 to 25] | 23 [18 to 29.5]
  AST, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  AST, Dose 2, Day 60 | 21 [18 to 26] | 21.5 [18 to 28.5]

51. Secondary Outcome: Levels of Basophils in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included basophil levels. Basophil levels were expressed in billion cells per liter (billion cells/L). Basophil levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Basophils, Dose 1, Day 0 | 0.03 [0.02 to 0.04] | 0.02 [0.02 to 0.03]
  Basophils, Dose 1 (Day 0 H6) | 0.03 [0.02 to 0.04] | 0.03 [0.02 to 0.03]
  Basophils, Dose 1 (Day 0 H12) | 0.03 [0.02 to 0.05] | 0.02 [0.02 to 0.03]
  Basophils, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Basophils, Dose 1 (Day 0 H18) | 0.03 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  Basophils, Dose 1, Day 1 | 0.03 [0.01 to 0.04] | 0.02 [0.02 to 0.03]
  Basophils, Dose 1, Day 7 | 0.03 [0.02 to 0.04] | 0.03 [0.02 to 0.04]
  Basophils, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Basophils, Dose 2, Day 30 | 0.03 [0.02 to 0.04] | 0.02 [0.02 to 0.04]
  Basophils, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Basophils, Dose 2 (Day 30 H6) | 0.03 [0.02 to 0.04] | 0.02 [0.02 to 0.03]
  Basophils, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Basophils, Dose 2 (Day 30 H12) | 0.02 [0.01 to 0.03] | 0.02 [0.02 to 0.04]
  Basophils, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Basophils, Dose 2 (Day 30 H18) | 0.03 [0.01 to 0.03] | 0.02 [0.01 to 0.03]
  Basophils, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Basophils, Dose 2, Day 31 | 0.02 [0.01 to 0.03] | 0.03 [0.02 to 0.04]
  Basophils, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Basophils, Dose 2, Day 37 | 0.03 [0.02 to 0.06] | 0.03 [0.02 to 0.03]
  Basophils, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Basophils, Dose 2, Day 60 | 0.03 [0.02 to 0.04] | 0.03 [0.02 to 0.03]

52. Secondary Outcome: Levels of Total Bilirubin in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included total bilirubin levels. Bilirubin concentrations were expressed in milligrams per deciliter (mG/dL). Bilirubin levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
mg/dL
  Total bilirubin, Dose 1, Day 0 | 0.5 [0.4 to 0.7] | 0.5 [0.3 to 0.7]
  Total bilirubin, Dose 1 (Day 0 H6) | 0.4 [0.25 to 0.5] | 0.4 [0.3 to 0.5]
  Total bilirubin, Dose 1 (Day 0 H12) | 0.4 [0.3 to 0.6] | 0.3 [0.3 to 0.5]
  Total bilirubin, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Total bilirubin, Dose 1 (Day 0 H18) | 0.6 [0.4 to 0.8] | 0.5 [0.3 to 0.6]
  Total bilirubin, Dose 1, Day 1 | 0.7 [0.6 to 0.9] | 0.5 [0.3 to 0.8]
  Total bilirubin, Dose 1, Day 7 | 0.5 [0.4 to 0.7] | 0.5 [0.3 to 0.6]
  Total bilirubin, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Total bilirubin, Dose 2, Day 30 | 0.6 [0.4 to 0.7] | 0.5 [0.4 to 0.7]
  Total bilirubin, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Total bilirubin, Dose 2 (Day 30 H6) | 0.4 [0.3 to 0.5] | 0.4 [0.3 to 0.5]
  Total bilirubin, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Total bilirubin, Dose 2 (Day 30 H12) | 0.5 [0.4 to 0.6] | 0.4 [0.3 to 0.5]
  Total bilirubin, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Total bilirubin, Dose 2 (Day 30 H18) | 0.6 [0.4 to 0.7] | 0.45 [0.3 to 0.5]
  Total bilirubin, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Total bilirubin, Dose 2, Day 31 | 0.7 [0.5 to 1] | 0.5 [0.45 to 0.7]
  Total bilirubin, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Total bilirubin, Dose 2, Day 37 | 0.5 [0.3 to 0.8] | 0.5 [0.4 to 0.65]
  Total bilirubin, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Total bilirubin, Dose 2, Day 60 | 0.5 [0.4 to 0.6] | 0.5 [0.4 to 0.6]

53. Secondary Outcome: Levels of Serum Creatinine in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included creatinine levels. Creatinine concentrations were expressed in milligrams per deciliter (mg/dL). Creatinine levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
mg/dL
  Creatinine, Dose 1, Day 0 | 0.8 [0.75 to 0.93] | 0.79 [0.72 to 0.85]
  Creatinine, Dose 1 (Day 0 H6) | 0.75 [0.66 to 0.85] | 0.72 [0.69 to 0.82]
  Creatinine, Dose 1 (Day 0 H12) | 0.78 [0.66 to 0.83] | 0.73 [0.68 to 0.83]
  Creatinine, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Creatinine, Dose 1 (Day 0 H18) | 0.7 [0.61 to 0.77] | 0.71 [0.63 to 0.84]
  Creatinine, Dose 1, Day 1 | 0.74 [0.68 to 0.91] | 0.77 [0.71 to 0.85]
  Creatinine, Dose 1, Day 7 | 0.81 [0.71 to 0.93] | 0.76 [0.69 to 0.87]
  Creatinine, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Creatinine, Dose 2, Day 30 | 0.82 [0.74 to 0.96] | 0.79 [0.72 to 0.83]
  Creatinine, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Creatinine, Dose 2 (Day 30 H6) | 0.75 [0.68 to 0.85] | 0.73 [0.67 to 0.83]
  Creatinine, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Creatinine, Dose 2 (Day 30 H12) | 0.76 [0.68 to 0.85] | 0.72 [0.69 to 0.82]
  Creatinine, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Creatinine, Dose 2 (Day 30 H18) | 0.74 [0.68 to 0.81] | 0.73 [0.65 to 0.82]
  Creatinine, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Creatinine, Dose 2, Day 31 | 0.79 [0.69 to 0.93] | 0.76 [0.7 to 0.87]
  Creatinine, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Creatinine, Dose 2, Day 37 | 0.81 [0.73 to 0.93] | 0.73 [0.7 to 0.9]
  Creatinine, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Creatinine, Dose 2, Day 60 | 0.84 [0.69 to 0.97] | 0.78 [0.72 to 0.91]

54. Secondary Outcome: Levels of Creatinine Phosphokinase (CPK) in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included CPK levels. CPK concentrations were expressed in milligrams per deciliter (mg/dL). CPK levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
mg/dL
  CPK, Dose 1, Day 0 | 75 [56.5 to 108] | 80 [62 to 148]
  CPK, Dose 1 (Day 0 H6 | 69.5 [53 to 106] | 75 [60 to 120]
  CPK, Dose 1 (Day 0 H12) | 64.5 [51 to 94.5] | 77 [57 to 110]
  CPK, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  CPK, Dose 1 (Day 0 H18) | 59 [49 to 90] | 61 [44 to 103]
  CPK, Dose 1, Day 1 | 54 [42.5 to 79.5] | 69 [46 to 96]
  CPK, Dose 1, Day 7 | 66 [55.5 to 95] | 80 [57 to 117]
  CPK, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  CPK, Dose 2, Day 30 | 83 [48 to 122] | 87 [55 to 145]
  CPK, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  CPK, Dose 2 (Day 30 H6) | 81 [45 to 108] | 86 [53.5 to 140.5]
  CPK, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  CPK, Dose 2 (Day 30 H12) | 72 [50 to 98] | 80.5 [54 to 134]
  CPK, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  CPK, Dose 2 (Day 30 H18) | 68.5 [53 to 103] | 70 [37 to 120]
  CPK, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  CPK, Dose 2, Day 31 | 67 [44 to 87] | 75 [50 to 119]
  CPK, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  CPK, Dose 2, Day 37 | 83 [59 to 119] | 93.5 [54 to 115.5]
  CPK, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  CPK, Dose 2, Day 60 | 82 [55 to 118] | 82.5 [62 to 122]

55. Secondary Outcome: Levels of C-reactive Protein (CRP) in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included CRP levels. CRP concentrations were expressed in milligrams per liter (mg/L). CRP levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
mg/L
  CRP, Dose 1, Day 0 | 1.15 [0.5 to 3] | 1.7 [0.5 to 2.5]
  CRP, Dose 1 (Day 0 H6) | 0.8 [0.5 to 2.9] | 1.6 [0.5 to 2.4]
  CRP, Dose 1 (Day 0 H12) | 1.5 [0.5 to 3.35] | 1.4 [0.5 to 2.1]
  CRP, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  CRP, Dose 1 (Day 0 H18) | 2.9 [1.5 to 4.4] | 1.25 [0.5 to 1.8]
  CRP, Dose 1, Day 1 | 5.8 [3.1 to 11.1] | 1.2 [0.5 to 1.8]
  CRP, Dose 1, Day 7 | 1.9 [0.5 to 4.25] | 1.3 [0.5 to 2.6]
  CRP, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  CRP, Dose 2, Day 30 | 1.3 [0.5 to 4.3] | 1.4 [0.5 to 3.1]
  CRP, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  CRP, Dose 2 (Day 30 H6) | 1.2 [0.5 to 2.3] | 1.5 [0.5 to 3.05]
  CRP, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  CRP, Dose 2 (Day 30 H12) | 1.8 [0.5 to 2.8] | 1.55 [0.5 to 3.1]
  CRP, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  CRP, Dose 2 (Day 30 H18) | 3.15 [2.1 to 5.3] | 0.75 [0.5 to 2.8]
  CRP, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  CRP, Dose 2, Day 31 | 5.8 [2.6 to 14.5] | 1.2 [0.5 to 2.65]
  CRP, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  CRP, Dose 2, Day 37 | 2.1 [1.1 to 5.8] | 1.3 [0.5 to 2.95]
  CRP, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  CRP, Dose 2, Day 60 | 1.4 [0.5 to 3.9] | 1.05 [0.5 to 3.85]

56. Secondary Outcome: Levels of Eosinophils in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included eosinophil levels. Eosinophil levels were expressed in billion cells per liter (billion cells/L). Eosinophil levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Eosinophils, Dose 1, Day 0 | 0.2 [0.11 to 0.25] | 0.13 [0.1 to 0.21]
  Eosinophils, Dose 1 (Day 0 H6) | 0.19 [0.13 to 0.27] | 0.13 [0.09 to 0.21]
  Eosinophils, Dose 1 (Day 0 H12) | 0.21 [0.15 to 0.27] | 0.17 [0.12 to 0.21]
  Eosinophils, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Eosinophils, Dose 1 (Day 0 H18) | 0.16 [0.12 to 0.3] | 0.2 [0.16 to 0.31]
  Eosinophils, Dose 1, Day 1 | 0.15 [0.08 to 0.25] | 0.1 [0.07 to 0.2]
  Eosinophils, Dose 1, Day 7 | 0.14 [0.08 to 0.2] | 0.11 [0.09 to 0.17]
  Eosinophils, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Eosinophils, Dose 2, Day 30 | 0.18 [0.11 to 0.25] | 0.14 [0.09 to 0.26]
  Eosinophils, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Eosinophils, Dose 2 (Day 30 H6) | 0.18 [0.1 to 0.29] | 0.13 [0.09 to 0.22]
  Eosinophils, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Eosinophils, Dose 2 (Day 30 H12) | 0.19 [0.12 to 0.31] | 0.14 [0.09 to 0.24]
  Eosinophils, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Eosinophils, Dose 2 (Day 30 H18) | 0.14 [0.05 to 0.21] | 0.19 [0.12 to 0.32]
  Eosinophils, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Eosinophils, Dose 2, Day 31 | 0.14 [0.05 to 0.2] | 0.13 [0.09 to 0.22]
  Eosinophils, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Eosinophils, Dose 2, Day 37 | 0.19 [0.11 to 0.24] | 0.15 [0.09 to 0.23]
  Eosinophils, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Eosinophils, Dose 2, Day 60 | 0.19 [0.1 to 0.28] | 0.14 [0.11 to 0.24]

57. Secondary Outcome: Levels of Haemoglobin in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included haemoglobin levels, expressed in grams per deciliter (g/dL). Haemoglobin levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: g/dL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
g/dL
  Haemoglobin, Dose 1, Day 0 | 13.35 [12.7 to 14.5] | 13.8 [12.5 to 14.8]
  Haemoglobin, Dose 1 (Day 0 H6) | 13.45 [12.3 to 14.05] | 13.6 [12.5 to 14.6]
  Haemoglobin, Dose 1 (Day 0 H12) | 13.25 [12.3 to 14.3] | 13.2 [12.6 to 14.5]
  Haemoglobin, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Haemoglobin, Dose 1 (Day 0 H18) | 12.6 [12 to 13.9] | 13.15 [12.5 to 14.5]
  Haemoglobin, Dose 1, Day 1 | 13.5 [12.6 to 14.45] | 13.8 [12.9 to 14.7]
  Haemoglobin, Dose 1, Day 7 | 13.35 [12.55 to 14.35] | 13.8 [12.8 to 14.6]
  Haemoglobin, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Haemoglobin, Dose 2, Day 30 | 13.7 [12.7 to 14.3] | 13.4 [12.6 to 14.3]
  Haemoglobin, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Haemoglobin, Dose 2 (Day 30 H6) | 13.4 [12.5 to 14] | 13.55 [12.45 to 14.15]
  Haemoglobin, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Haemoglobin, Dose 2 (Day 30 H12) | 13.2 [12.6 to 14.1] | 13.1 [12.4 to 14.15]
  Haemoglobin, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Haemoglobin, Dose 2 (Day 30 H18) | 13.15 [11.7 to 13.9] | 13.05 [12.3 to 14.1]
  Haemoglobin, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Haemoglobin, Dose 2, Day 31 | 13.5 [12.5 to 14.4] | 13.75 [12.65 to 14.6]
  Haemoglobin, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Haemoglobin, Dose 2, Day 37 | 13.6 [12.6 to 14.5] | 13.65 [12.35 to 14.5]
  Haemoglobin, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Haemoglobin, Dose 2, Day 60 | 13.5 [12.4 to 14.5] | 13.8 [12.2 to 14.5]

58. Secondary Outcome: Levels of Lactate Dehydrogenase (LDH) in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included LDH levels, expressed in units per liter (U/L). LDH levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
U/L
  LDH, Dose 1, Day 0 | 401.5 [377 to 473.5] | 382 [346 to 438]
  LDH, Dose 1 (Day 0 H6) | 414 [388.5 to 449.5] | 389 [353 to 423]
  LDH, Dose 1 (Day 0 H12) | 412 [392 to 457.5] | 378 [339 to 426]
  LDH, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  LDH, Dose 1 (Day 0 H18) | 422 [341 to 461] | 369.5 [302 to 410]
  LDH, Dose 1, Day 1 | 389 [352 to 466] | 367 [342 to 411]
  LDH, Dose 1, Day 7 | 417.5 [382.5 to 479.5] | 392 [371 to 436]
  LDH, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  LDH, Dose 2, Day 30 | 391 [360 to 456] | 395 [348 to 426]
  LDH, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  LDH, Dose 2 (Day 30 H6) | 437 [397 to 470] | 396.5 [350.5 to 428]
  LDH, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  LDH, Dose 2 (Day 30 H12) | 425 [403 to 470] | 382.5 [338.5 to 424]
  LDH, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  LDH, Dose 2 (Day 30 H18) | 403 [365 to 450] | 334.5 [297 to 390]
  LDH, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  LDH, Dose 2, Day 31 | 408 [373 to 453] | 372 [354 to 403]
  LDH, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  LDH, Dose 2, Day 37 | 442 [412 to 464] | 403 [368.5 to 446]
  LDH, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  LDH, Dose 2, Day 60 | 422 [397 to 478] | 404 [374 to 431.5]

59. Secondary Outcome: Levels of Lymphocytes in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included lymphocyte levels. Lymphocyte levels were expressed in billion cells per liter (billion cells/L). Lymphocyte levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Lymphocytes, Dose 1, Day 0 | 1.84 [1.45 to 1.98] | 1.99 [1.61 to 2.26]
  Lymphocytes, Dose 1 (Day 0 H6) | 1.89 [1.48 to 2.35] | 2.07 [1.52 to 2.46]
  Lymphocytes, Dose 1 (Day 0 H12) | 1.97 [1.72 to 2.33] | 2.39 [2 to 2.97]
  Lymphocytes, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Lymphocytes, Dose 1 (Day 0 H18) | 1.73 [1.41 to 2.48] | 3.08 [2.45 to 3.53]
  Lymphocytes, Dose 1, Day 1 | 1.58 [1.25 to 1.83] | 1.94 [1.66 to 2.26]
  Lymphocytes, Dose 1, Day 7 | 1.69 [1.37 to 1.91] | 1.97 [1.56 to 2.17]
  Lymphocytes, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Lymphocytes, Dose 2, Day 30 | 1.67 [1.36 to 2.03] | 1.97 [1.64 to 2.5]
  Lymphocytes, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Lymphocytes, Dose 2 (Day 30 H6) | 1.81 [1.56 to 2.16] | 2.11 [1.78 to 2.59]
  Lymphocytes, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Lymphocytes, Dose 2 (Day 30 H12) | 1.9 [1.36 to 2.39] | 2.35 [2.1 to 2.82]
  Lymphocytes, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Lymphocytes, Dose 2 (Day 30 H18) | 1.46 [1.06 to 1.83] | 2.99 [2.45 to 3.53]
  Lymphocytes, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Lymphocytes, Dose 2, Day 31 | 1.19 [0.89 to 1.43] | 2.01 [1.75 to 2.5]
  Lymphocytes, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Lymphocytes, Dose 2, Day 37 | 1.74 [1.41 to 2.21] | 2.01 [1.64 to 2.36]
  Lymphocytes, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Lymphocytes, Dose 2, Day 60 | 1.76 [1.4 to 2.29] | 2.09 [1.73 to 2.31]

60. Secondary Outcome: Levels of Monocytes in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included monocyte levels. Monocyte levels were expressed in billion cells per liter (billion cells/L). Monocyte levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Monocytes, Dose 1, Day 0 | 0.55 [0.45 to 0.66] | 0.55 [0.4 to 0.62]
  Monocytes, Dose 1 (Day 0 H6) | 0.67 [0.59 to 0.76] | 0.52 [0.4 to 0.55]
  Monocytes, Dose 1 (Day 0 H12) | 0.79 [0.62 to 0.9] | 0.53 [0.41 to 0.6]
  Monocytes, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Monocytes, Dose 1 (Day 0 H18) | 0.79 [0.66 to 0.92] | 0.59 [0.5 to 0.61]
  Monocytes, Dose 1, Day 1 | 0.72 [0.6 to 0.84] | 0.45 [0.4 to 0.54]
  Monocytes, Dose 1, Day 7 | 0.54 [0.43 to 0.63] | 0.44 [0.37 to 0.58]
  Monocytes, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Monocytes, Dose 2, Day 30 | 0.55 [0.47 to 0.65] | 0.5 [0.43 to 0.63]
  Monocytes, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Monocytes, Dose 2 (Day 30 H6) | 0.67 [0.54 to 0.78] | 0.48 [0.4 to 0.56]
  Monocytes, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Monocytes, Dose 2 (Day 30 H12) | 0.66 [0.57 to 0.87] | 0.51 [0.39 to 0.61]
  Monocytes, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Monocytes, Dose 2 (Day 30 H18) | 0.8 [0.62 to 0.94] | 0.49 [0.43 to 0.59]
  Monocytes, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Monocytes, Dose 2, Day 31 | 0.67 [0.53 to 0.81] | 0.51 [0.44 to 0.67]
  Monocytes, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Monocytes, Dose 2, Day 37 | 0.51 [0.39 to 0.64] | 0.51 [0.44 to 0.59]
  Monocytes, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Monocytes, Dose 2, Day 60 | 0.51 [0.39 to 0.68] | 0.52 [0.44 to 0.64]

61. Secondary Outcome: Levels of Neutrophils in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included neutrophil levels. Neutrophil levels were expressed in billion cells per liter (billion cells/L). Neutrophil levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Neutrophils, Dose 1, Day 0 | 3.7 [3 to 5.49] | 3.36 [2.77 to 4.21]
  Neutrophils, Dose 1 (Day 0 H6) | 6.48 [5.02 to 7.84] | 4.12 [2.96 to 4.41]
  Neutrophils, Dose 1 (Day 0 H12) | 7.61 [6.87 to 9.01] | 3.39 [3 to 4.53]
  Neutrophils, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Neutrophils, Dose 1 (Day 0 H18) | 6.07 [5.56 to 8.31] | 3.61 [3.31 to 4.12]
  Neutrophils, Dose 1, Day 1 | 6.13 [4.26 to 6.76] | 3.76 [3.12 to 4.23]
  Neutrophils, Dose 1, Day 7 | 4.17 [3.05 to 5.17] | 3.46 [2.73 to 4.19]
  Neutrophils, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Neutrophils, Dose 2, Day 30 | 3.66 [3.08 to 4.49] | 2.91 [2.43 to 3.91]
  Neutrophils, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Neutrophils, Dose 2 (Day 30 H6) | 5.9 [5.28 to 7.75] | 3.39 [2.93 to 4.07]
  Neutrophils, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Neutrophils, Dose 2 (Day 30 H12) | 7.07 [6.47 to 8.58] | 3.36 [2.59 to 4.12]
  Neutrophils, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Neutrophils, Dose 2 (Day 30 H18) | 7.42 [6.84 to 9.35] | 3.02 [2.39 to 3.74]
  Neutrophils, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Neutrophils, Dose 2, Day 31 | 6.32 [4.78 to 7.41] | 3.2 [2.77 to 4.9]
  Neutrophils, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Neutrophils, Dose 2, Day 37 | 3.64 [2.73 to 5.48] | 3.13 [2.68 to 4.47]
  Neutrophils, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Neutrophils, Dose 2, Day 60 | 3.96 [3.16 to 4.96] | 2.95 [2.5 to 3.71]

62. Secondary Outcome: Platelet Count in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included platelet count levels. Platelet count levels were expressed in billion cells per liter (billion cells/L). Platelet count levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  Platelets, Dose 1, Day 0 | 228 [191.5 to 261.5] | 225 [207 to 266]
  Platelets, Dose 1 (Day 0 H6) | 229 [204 to 259.5] | 231 [212 to 263]
  Platelets, Dose 1 (Day 0 H12) | 235 [193 to 259] | 230 [217 to 263]
  Platelets, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Platelets, Dose 1 (Day 0 H18) | 222 [186 to 260] | 233 [215 to 274]
  Platelets, Dose 1, Day 1 | 220.5 [187.5 to 258] | 227 [206 to 269]
  Platelets, Dose 1, Day 7 | 263.5 [215.5 to 291] | 247 [217 to 268]
  Platelets, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Platelets, Dose 2, Day 30 | 224 [185 to 267] | 228 [204 to 260]
  Platelets, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Platelets, Dose 2 (Day 30 H6) | 238 [195 to 270] | 232 [212 to 261.5]
  Platelets, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Platelets, Dose 2 (Day 30 H12) | 226 [194 to 260] | 234 [213.5 to 258]
  Platelets, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Platelets, Dose 2 (Day 30 H18) | 230.5 [179 to 276] | 229 [199 to 275]
  Platelets, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Platelets, Dose 2, Day 31 | 218 [170 to 238] | 217.5 [204.5 to 256.5]
  Platelets, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Platelets, Dose 2, Day 37 | 253 [205 to 301] | 243 [208.5 to 282]
  Platelets, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Platelets, Dose 2, Day 60 | 240 [195 to 283] | 241.5 [208 to 276.5]

63. Secondary Outcome: Levels of Red Blood Cell (RBC) in Blood Samples - Step 1
Description: Haematological laboratory parameters assessed included red blood cells levels, expressed in trillion cells per liter (trillion cells/L). RBC levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: trillion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
trillion cells/L
  RBC, Dose 1, Day 0 | 4.51 [4.33 to 4.83] | 4.56 [4.27 to 4.96]
  RBC, Dose 1 (Day 0 H6) | 4.45 [4.18 to 4.82] | 4.58 [4.24 to 4.78]
  RBC, Dose 1 (Day 0 H12) | 4.42 [4.12 to 4.68] | 4.51 [4.27 to 4.78]
  RBC, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  RBC, Dose 1 (Day 0 H18) | 4.19 [4.02 to 4.79] | 4.36 [4.19 to 4.72]
  RBC, Dose 1, Day 1 | 4.48 [4.25 to 4.85] | 4.62 [4.36 to 4.78]
  RBC, Dose 1, Day 7 | 4.54 [4.24 to 4.75] | 4.54 [4.38 to 4.92]
  RBC, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  RBC, Dose 2, Day 30 | 4.48 [4.27 to 4.7] | 4.53 [4.25 to 4.79]
  RBC, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  RBC, Dose 2 (Day 30 H6) | 4.43 [4.14 to 4.6] | 4.49 [4.26 to 4.8]
  RBC, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  RBC, Dose 2 (Day 30 H12) | 4.33 [4.21 to 4.62] | 4.46 [4.25 to 4.71]
  RBC, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  RBC, Dose 2 (Day 30 H18) | 4.22 [3.86 to 4.66] | 4.34 [4.09 to 4.62]
  RBC, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  RBC, Dose 2, Day 31 | 4.42 [4.12 to 4.85] | 4.58 [4.38 to 4.9]
  RBC, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  RBC, Dose 2, Day 37 | 4.5 [4.13 to 4.84] | 4.52 [4.2 to 4.88]
  RBC, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  RBC, Dose 2, Day 60 | 4.5 [4.14 to 4.94] | 4.61 [4.41 to 4.85]

64. Secondary Outcome: Levels of Urea in Blood Samples - Step 1
Description: Biochemical laboratory parameters assessed included urea levels, expressed in miligrams per deciliter (mg/dL). Urea levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
mg/dL
  Urea Nitrogen, Dose 1, Day 0 | 27.5 [23 to 35.5] | 30 [26 to 35]
  Urea Nitrogen, Dose 1 (Day 0 H6) | 27 [24 to 31.5] | 30 [26 to 34]
  Urea Nitrogen, Dose 1 (Day 0 H12) | 27 [24 to 31.5] | 29 [27 to 32]
  Urea Nitrogen, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  Urea Nitrogen, Dose 1 (Day 0 H18) | 23 [21 to 32] | 27 [24 to 30]
  Urea Nitrogen, Dose 1, Day 1 | 23.5 [18.5 to 29] | 25 [23 to 30]
  Urea Nitrogen, Dose 1, Day 7 | 27.5 [24.5 to 35] | 27 [23 to 31]
  Urea Nitrogen, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  Urea Nitrogen, Dose 2, Day 30 | 28 [25 to 37] | 26 [22 to 33]
  Urea Nitrogen, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  Urea Nitrogen, Dose 2 (Day 30 H6) | 29 [24 to 34] | 26 [23 to 32.5]
  Urea Nitrogen, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  Urea Nitrogen, Dose 2 (Day 30 H12) | 28 [24 to 34] | 27 [23.5 to 32]
  Urea Nitrogen, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  Urea Nitrogen, Dose 2 (Day 30 H18) | 25.5 [21 to 31] | 24.5 [22 to 28]
  Urea Nitrogen, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  Urea Nitrogen, Dose 2, Day 31 | 23 [19 to 30] | 26 [21 to 28.5]
  Urea Nitrogen, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  Urea Nitrogen, Dose 2, Day 37 | 26 [22 to 36] | 25.5 [23 to 31]
  Urea Nitrogen, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  Urea Nitrogen, Dose 2, Day 60 | 29 [22 to 33] | 27 [23.5 to 30]

65. Secondary Outcome: Levels of White Blood Cells (WBC) - Step 1
Description: Haematological laboratory parameters assessed included WBC levels. WBC levels were expressed in billion cells per liter (billion cells/L). WBC levels were assessed at different time points (plus 6, 12 and 18 hours - H6, H12, H18) on Day 0 and Day 30.
Time Frame: as for outcome 49
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 28 | 29
billion cells/L
  WBC, Dose 1, Day 0 | 6.25 [5.53 to 8.49] | 6.33 [5.46 to 7.03]
  WBC, Dose 1 (Day 0 H6) | 9.73 [7.7 to 11.3] | 6.49 [5.78 to 7.37]
  WBC, Dose 1 (Day 0 H12) | 10.45 [9.75 to 12.4] | 6.84 [6 to 7.4]
  WBC, Dose 1 (Day 0 H18): number analyzed (Participants) | 15 | 14
  WBC, Dose 1 (Day 0 H18) | 8.72 [7.63 to 12.2] | 7.43 [7.15 to 8.02]
  WBC, Dose 1, Day 1 | 8.7 [6.37 to 9.7] | 6.25 [5.85 to 6.83]
  WBC, Dose 1, Day 7 | 6.67 [5.49 to 8.17] | 6.14 [5.27 to 7.32]
  WBC, Dose 2, Day 30: number analyzed (Participants) | 27 | 27
  WBC, Dose 2, Day 30 | 6.04 [5.48 to 8.07] | 5.77 [4.96 to 7.21]
  WBC, Dose 2 (Day 30 H6): number analyzed (Participants) | 27 | 28
  WBC, Dose 2 (Day 30 H6) | 9.28 [7.91 to 10.4] | 6.07 [5.76 to 6.96]
  WBC, Dose 2 (Day 30 H12): number analyzed (Participants) | 27 | 28
  WBC, Dose 2 (Day 30 H12) | 9.88 [9.29 to 11.4] | 6.28 [5.8 to 7.37]
  WBC, Dose 2 (Day 30 H18): number analyzed (Participants) | 14 | 14
  WBC, Dose 2 (Day 30 H18) | 9.57 [8.24 to 12.2] | 6.8 [6.49 to 7.21]
  WBC, Dose 2, Day 31: number analyzed (Participants) | 27 | 28
  WBC, Dose 2, Day 31 | 8.21 [6.78 to 9.36] | 6.34 [5.67 to 7.16]
  WBC, Dose 2, Day 37: number analyzed (Participants) | 27 | 28
  WBC, Dose 2, Day 37 | 5.7 [5.13 to 8.46] | 6.25 [5.46 to 7.31]
  WBC, Dose 2, Day 60: number analyzed (Participants) | 27 | 28
  WBC, Dose 2, Day 60 | 6.48 [5.45 to 8.24] | 6.07 [5.04 to 6.7]

66. Secondary Outcome: Levels of Diastolic Blood Pressure - Step 1
Description: Diastolic pressure was part of the list of vital signs followed at specific protocol-defined time points during this study, measured in millimeter of mercury (mmHg). On Days -30, 0 and 30, diastolic blood pressure was assessed at multiple time points (plus 1.5, 3, 6, 9, 12 and 18 hours - H1.5, H3, H6, H9, H12 and H18).
Time Frame: At Day -30, -30 (H1.5, H3, H6, H9, H12, H18) -29, - 28, - 27, -23, 0, 0 (H1.5, H6, H12 H18), 1, 2, 7, 30, 30 (H1.5, H3, H6, H9, H12, H18), 31, 32, 33, 37 and 60
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
mmHg
  Diastolic, placebo (D-30) | 81 [74 to 86] | 76.5 [67 to 83]
  Diastolic, placebo (D-30 H1.5) | 75 [69 to 83] | 72 [65 to 79]
  Diastolic, placebo (D-30 H3) | 75.5 [68 to 83] | 71.5 [65 to 80]
  Diastolic, placebo (D-30 H6) | 73.5 [67 to 83] | 71.5 [67 to 82]
  Diastolic, placebo (D-30 H9) | 76 [71 to 86] | 75 [67 to 84]
  Diastolic, placebo (D-30 H12) | 78 [69 to 84] | 72.5 [66 to 80]
  Diastolic, placebo (D-30 H18): number analyzed (Participants) | 15 | 15
  Diastolic, placebo (D-30 H18) | 75 [67 to 80] | 68 [64 to 84]
  Diastolic, placebo (D-29) | 77 [70 to 83] | 73.5 [64 to 81]
  Diastolic, placebo (D-28): number analyzed (Participants) | 29 | 30
  Diastolic, placebo (D-28) | 75 [70 to 83] | 74.5 [69 to 78]
  Diastolic, placebo (D-27): number analyzed (Participants) | 29 | 30
  Diastolic, placebo (D-27) | 78 [72 to 82] | 75 [71 to 81]
  Diastolic, placebo (D-23): number analyzed (Participants) | 29 | 30
  Diastolic, placebo (D-23) | 76 [71 to 81] | 75.5 [66 to 80]
  Diastolic, Dose 1 (D0): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D0) | 76 [70.5 to 83] | 76 [68 to 85]
  Diastolic, Dose 1 (D0 H1.5): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D0 H1.5) | 74 [70 to 81] | 73 [67 to 78]
  Diastolic, Dose 1 (D0 H6): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D0 H6) | 73.5 [67.5 to 80] | 72 [65 to 78]
  Diastolic, Dose 1 (D0 H12): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D0 H12) | 72 [69 to 79.5] | 72 [66 to 79]
  Diastolic, Dose 1 (D0 H18): number analyzed (Participants) | 15 | 14
  Diastolic, Dose 1 (D0 H18) | 73 [61 to 78] | 66.5 [60 to 78]
  Diastolic, Dose 1 (D1): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D1) | 72 [69 to 79] | 76 [66 to 80]
  Diastolic, Dose 1 (D2): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D2) | 74 [70 to 81.5] | 73 [67 to 79]
  Diastolic, Dose 1 (D7): number analyzed (Participants) | 28 | 29
  Diastolic, Dose 1 (D7) | 75 [71 to 79.5] | 73 [70 to 82]
  Diastolic, Dose 2 (D30): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30) | 76 [69 to 80] | 77.5 [68.5 to 83]
  Diastolic, Dose 2 (D30 H1.5): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30 H1.5) | 72 [67 to 78] | 70 [66 to 76.5]
  Diastolic, Dose 2 (D30 H3): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30 H3) | 72 [68 to 79] | 72 [63 to 78]
  Diastolic, Dose 2 (D30 H6): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30 H6) | 72 [69 to 75] | 70.5 [65.5 to 75.5]
  Diastolic, Dose 2 (D30 H9): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30 H9) | 75 [71 to 79] | 75 [65.5 to 81.5]
  Diastolic, Dose 2 (D30 H12): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D30 H12) | 73 [68 to 78] | 72.5 [66.5 to 79.5]
  Diastolic, Dose 2 (D30 H18): number analyzed (Participants) | 14 | 14
  Diastolic, Dose 2 (D30 H18) | 70 [64 to 74] | 71.5 [66 to 79]
  Diastolic, Dose 2 (D31): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D31) | 71 [67 to 77] | 71 [65.5 to 80]
  Diastolic, Dose 2 (D32): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D32) | 77 [71 to 81] | 74 [67 to 79]
  Diastolic, Dose 2 (D33): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D33) | 77 [71 to 81] | 73 [70.5 to 79.5]
  Diastolic, Dose 2 (D37): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D37) | 76 [68 to 86] | 74 [68.5 to 79.5]
  Diastolic, Dose 2 (D60): number analyzed (Participants) | 27 | 28
  Diastolic, Dose 2 (D60) | 78 [72 to 84] | 73 [67 to 81.5]

67. Secondary Outcome: Levels of Heart Rate - Step 1
Description: Heart rate was part of the list of vital signs followed at specific protocol-defined timepoints during this study. It was expressed in beats per minute. On Days -30, 0 and 30, heart rate was assessed at multiple time points (plus 1.5, 3, 6, 9, 12 and 18 hours - H1.5, H3, H6, H9, H12 and H18).
Time Frame: as for outcome 66
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: beats/minute
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
beats/minute
  Heart rate, placebo (D-30) | 75.5 [62 to 86] | 70 [64 to 79]
  Heart rate, placebo (D-30 H1.5) | 75 [62 to 82] | 73 [62 to 77]
  Heart rate, placebo (D-30 H3) | 69.5 [56 to 76] | 63.5 [58 to 71]
  Heart rate, placebo (D-30 H6) | 69 [61 to 78] | 69 [60 to 80]
  Heart rate, placebo (D-30 H9) | 66.5 [56 to 82] | 65 [55 to 70]
  Heart rate, placebo (D-30 H12) | 71.5 [64 to 80] | 72.5 [60 to 81]
  Heart rate, placebo (D-30 H18): number analyzed (Participants) | 15 | 15
  Heart rate, placebo (D-30 H18) | 66 [55 to 75] | 70 [66 to 77]
  Heart rate, placebo (D-29) | 74.5 [63 to 82] | 65.5 [62 to 70]
  Heart rate, placebo (D-28): number analyzed (Participants) | 29 | 30
  Heart rate, placebo (D-28) | 70 [66 to 82] | 73.5 [65 to 81]
  Heart rate, placebo (D-27): number analyzed (Participants) | 29 | 30
  Heart rate, placebo (D-27) | 72 [66 to 80] | 70 [65 to 81]
  Heart rate, placebo (D-23): number analyzed (Participants) | 29 | 30
  Heart rate, placebo (D-23) | 72 [66 to 80] | 66 [58 to 75]
  Heart rate, Dose 1 (D0): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D0) | 69.5 [62 to 80.5] | 72 [62 to 79]
  Heart rate, Dose 1 (D0 H1.5): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D0 H1.5) | 67.5 [62 to 76] | 68 [62 to 77]
  Heart rate, Dose 1 (D0 H6): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D0 H6) | 66 [60.5 to 80.5] | 68 [65 to 79]
  Heart rate, Dose 1 (D0 H12): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D0 H12) | 76 [66.5 to 83] | 69 [61 to 79]
  Heart rate, Dose 1 (D0 H18): number analyzed (Participants) | 15 | 14
  Heart rate, Dose 1 (D0 H18) | 76 [60 to 83] | 67 [60 to 77]
  Heart rate, Dose 1 (D1): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D1) | 72 [65 to 82] | 67 [64 to 75]
  Heart rate, Dose 1 (D2): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D2) | 71.5 [60 to 80] | 69 [65 to 79]
  Heart rate, Dose 1 (D7): number analyzed (Participants) | 28 | 29
  Heart rate, Dose 1 (D7) | 74 [63 to 80.5] | 71 [62 to 82]
  Heart rate, Dose 2 (D30): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30) | 65 [59 to 77] | 66.5 [58 to 76.5]
  Heart rate, Dose 2 (D30 H1.5): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30 H1.5) | 69 [60 to 78] | 68.5 [57.5 to 79]
  Heart rate, Dose 2 (D30 H3): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30 H3) | 66 [55 to 74] | 65 [60.5 to 76]
  Heart rate, Dose 2 (D30 H6): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30 H6) | 73 [64 to 80] | 71.5 [62.5 to 81]
  Heart rate, Dose 2 (D30 H9): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30 H9) | 72 [57 to 81] | 65.5 [59 to 79]
  Heart rate, Dose 2 (D30 H12): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D30 H12) | 79 [66 to 85] | 69.5 [63 to 81]
  Heart rate, Dose 2 (D30 H18): number analyzed (Participants) | 14 | 14
  Heart rate, Dose 2 (D30 H18) | 84.5 [79 to 90] | 74.5 [66 to 80]
  Heart rate, Dose 2 (D31): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D31) | 81 [65 to 89] | 66.5 [58 to 77.5]
  Heart rate, Dose 2 (D32): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D32) | 70 [63 to 83] | 70.5 [62 to 77.5]
  Heart rate, Dose 2 (D33): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D33) | 69 [63 to 81] | 70.5 [64.5 to 79]
  Heart rate, Dose 2 (D37): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D37) | 67 [59 to 79] | 72.5 [61.5 to 79.5]
  Heart rate, Dose 2 (D60): number analyzed (Participants) | 27 | 28
  Heart rate, Dose 2 (D60) | 72 [67 to 80] | 71 [63.5 to 79.5]

68. Secondary Outcome: Levels of Respiratory Rate - Step 1
Description: Respiratory Rate was part of the list of vital signs followed at specific protocol-defined timepoints during this study. It was expressed as breaths per minute (breaths/min). On Days -30, 0 and 30, respiratory rate was assessed at multiple time points (plus 1.5, 3, 6, 9, 12 and 18 hours - H1.5, H3, H6, H9, H12 and H18).
Time Frame: as for outcome 66
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: breaths/min
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
breaths/min
  Respiratory Rate, placebo (D-30) | 14 [12 to 16] | 13 [12 to 16]
  Respiratory Rate, placebo (D-30 H1.5) | 13 [12 to 15] | 14.5 [13 to 16]
  Respiratory Rate, placebo (D-30 H3) | 13 [12 to 15] | 14 [12 to 15]
  Respiratory Rate, placebo (D-30 H6) | 12.5 [12 to 16] | 14 [13 to 16]
  Respiratory Rate, placebo (D-30 H9) | 13 [12 to 15] | 15 [13 to 16]
  Respiratory Rate, placebo (D-30 H12) | 14 [12 to 15] | 14.5 [13 to 15]
  Respiratory Rate, placebo (D-30 H18): number analyzed (Participants) | 15 | 15
  Respiratory Rate, placebo (D-30 H18) | 13 [12 to 14] | 12 [11 to 14]
  Respiratory Rate, placebo (D-29) | 13.5 [12 to 16] | 14 [13 to 15]
  Respiratory Rate, placebo (D-28): number analyzed (Participants) | 29 | 30
  Respiratory Rate, placebo (D-28) | 14 [12 to 16] | 14 [13 to 16]
  Respiratory Rate, placebo (D-27): number analyzed (Participants) | 29 | 30
  Respiratory Rate, placebo (D-27) | 14 [12 to 14] | 14 [13 to 14]
  Respiratory Rate, placebo (D-23): number analyzed (Participants) | 29 | 30
  Respiratory Rate, placebo (D-23) | 14 [12 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 1 (D0): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D0) | 14 [12.5 to 15.5] | 14 [12 to 15]
  Respiratory Rate, Dose 1 (D0 H1.5): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D0 H1.5) | 14 [12 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 1 (D0 H6): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D0 H6) | 14 [13 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 1 (D0 H12): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D0 H12) | 13.5 [12 to 14] | 14 [13 to 14]
  Respiratory Rate, Dose 1 (D0 H18): number analyzed (Participants) | 15 | 14
  Respiratory Rate, Dose 1 (D0 H18) | 13 [12 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 1 (D1): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D1) | 14 [12 to 15] | 14 [13 to 14]
  Respiratory Rate, Dose 1 (D2): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D2) | 14 [13 to 14.5] | 14 [12 to 15]
  Respiratory Rate, Dose 1 (D7): number analyzed (Participants) | 28 | 29
  Respiratory Rate, Dose 1 (D7) | 13.5 [13 to 14.5] | 13 [13 to 14]
  Respiratory Rate, Dose 2 (D30): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30) | 14 [12 to 15] | 14 [12 to 16]
  Respiratory Rate, Dose 2 (D30 H1.5): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30 H1.5) | 14 [13 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 2 (D30 H3): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30 H3) | 14 [12 to 15] | 14 [12 to 15]
  Respiratory Rate, Dose 2 (D30 H6): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30 H6) | 13 [12 to 15] | 14 [12 to 15]
  Respiratory Rate, Dose 2 (D30 H9): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30 H9) | 14 [12 to 15] | 13.5 [12.5 to 14]
  Respiratory Rate, Dose 2 (D30 H12): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D30 H12) | 14 [12 to 15] | 14 [13 to 15]
  Respiratory Rate, Dose 2 (D30 H18): number analyzed (Participants) | 14 | 14
  Respiratory Rate, Dose 2 (D30 H18) | 14 [12 to 15] | 14 [14 to 15]
  Respiratory Rate, Dose 2 (D31): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D31) | 13 [12 to 15] | 14 [12 to 15]
  Respiratory Rate, Dose 2 (D32): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D32) | 14 [12 to 14] | 14 [13 to 15]
  Respiratory Rate, Dose 2 (D33): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D33) | 13 [12 to 14] | 14 [13 to 15]
  Respiratory Rate, Dose 2 (D37): number analyzed (Participants) | 27 | 28
  Respiratory Rate, Dose 2 (D37) | 14 [12 to 16] | 14 [12.5 to 15]
  Respiratory Rate, Dose 2 (D60): number analyzed (Participants) | 25 | 26
  Respiratory Rate, Dose 2 (D60) | 14 [12 to 15] | 14 [13 to 16]

69. Secondary Outcome: Levels of Systolic Pressure - Step 1
Description: Systolic pressure was part of the list of vital signs followed at specific protocol-defined time points during this study, measured in millimeter of mercury (mmHg). On Days -30, 0 and 30, systolic pressure was assessed at multiple time points (plus 1.5, 3, 6, 9, 12 and 18 hours - H1.5, H3, H6, H9, H12 and H18).
Time Frame: as for outcome 66
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 30 | 30
mmHg
  Systolic, placebo (D-30) | 123.5 [112 to 130] | 116 [106 to 125]
  Systolic, placebo (D-30 H1.5) | 117 [111 to 124] | 114 [103 to 124]
  Systolic, placebo (D-30 H3) | 117.5 [112 to 126] | 114 [105 to 118]
  Systolic, placebo (D-30 H6) | 118 [113 to 124] | 112 [105 to 124]
  Systolic, placebo (D-30 H9) | 120.5 [112 to 131] | 114.5 [106 to 123]
  Systolic, placebo (D-30 H12) | 121.5 [112 to 129] | 112 [105 to 125]
  Systolic, placebo (D-30 H18): number analyzed (Participants) | 15 | 15
  Systolic, placebo (D-30 H18) | 111 [106 to 122] | 106 [96 to 118]
  Systolic, placebo (D-29) | 116.5 [111 to 124] | 112 [104 to 122]
  Systolic, placebo (D-28): number analyzed (Participants) | 29 | 30
  Systolic, placebo (D-28) | 121 [110 to 124] | 114 [103 to 121]
  Systolic, placebo (D-27): number analyzed (Participants) | 29 | 30
  Systolic, placebo (D-27) | 119 [112 to 124] | 115.5 [109 to 121]
  Systolic, placebo (D-23): number analyzed (Participants) | 29 | 30
  Systolic, placebo (D-23) | 118 [110 to 123] | 115 [104 to 122]
  Systolic, Dose 1 (D0): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D0) | 118 [112 to 122.5] | 114 [108 to 124]
  Systolic, Dose 1 (D0 H1.5): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D0 H1.5) | 116 [110.5 to 121.5] | 109 [102 to 119]
  Systolic, Dose 1 (D0 H6): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D0 H6) | 117 [111 to 121.5] | 112 [103 to 117]
  Systolic, Dose 1 (D0 H12): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D0 H12) | 115 [110 to 126] | 114 [107 to 120]
  Systolic, Dose 1 (D0 H18): number analyzed (Participants) | 15 | 14
  Systolic, Dose 1 (D0 H18) | 112 [104 to 121] | 105 [99 to 122]
  Systolic, Dose 1 (D1): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D1) | 114 [108.5 to 119] | 114 [104 to 123]
  Systolic, Dose 1 (D2): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D2) | 115 [110 to 124] | 111 [103 to 118]
  Systolic, Dose 1 (D7): number analyzed (Participants) | 28 | 29
  Systolic, Dose 1 (D7) | 116 [111 to 120.5] | 113 [107 to 123]
  Systolic, Dose 2 (D30): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30) | 115 [112 to 121] | 112.5 [106.5 to 122.5]
  Systolic, Dose 2 (D30 H1.5): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30 H1.5) | 115 [108 to 124] | 109.5 [102 to 117.5]
  Systolic, Dose 2 (D30 H3): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30 H3) | 116 [111 to 124] | 113 [103 to 120.5]
  Systolic, Dose 2 (D30 H6): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30 H6) | 117 [107 to 122] | 112 [103.5 to 118]
  Systolic, Dose 2 (D30 H9): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30 H9) | 117 [108 to 121] | 116 [108.5 to 124]
  Systolic, Dose 2 (D30 H12): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D30 H12) | 116 [109 to 125] | 116.5 [105 to 122]
  Systolic, Dose 2 (D30 H18): number analyzed (Participants) | 14 | 14
  Systolic, Dose 2 (D30 H18) | 109.5 [102 to 115] | 107 [100 to 122]
  Systolic, Dose 2 (D31): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D31) | 114 [108 to 123] | 109.5 [104 to 119]
  Systolic, Dose 2 (D32): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D32) | 116 [113 to 120] | 110.5 [103 to 115.5]
  Systolic, Dose 2 (D33): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D33) | 116 [112 to 122] | 111.5 [106 to 119.5]
  Systolic, Dose 2 (D37): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D37) | 120 [108 to 126] | 112 [106 to 124.5]
  Systolic, Dose 2 (D60): number analyzed (Participants) | 27 | 28
  Systolic, Dose 2 (D60) | 120 [109 to 125] | 115 [106.5 to 122.5]

70. Secondary Outcome: Anti-Hepatitis B Surface (Anti-HBs) Antibody Concentrations in Serum - Step 2 Immuno
Description: Anti-HBs antibody concentrations in serum were measured by CLIA Assay. Concentrations were presented as geometric mean concentrations, in milli-International Units per milliliter (mIU/mL).
Time Frame: At Day 0 (PRE) and post-vaccination (Day 44 for HBsAg/AS_2 Group and Day 194 for Engerix-B_2 Group)
Population: Analyses were performed on the According-To-Protocol (ATP) cohort for adaptive immunogenicity up to 30 days (step 2 only) post last vaccination, which included all evaluable subjects, who complied with the protocol and for whom data concerning adaptive immunogenicity were available for at least one adaptive assay at one post-vaccination time point.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 8
mIU/mL
  Anti-HBs, PRE | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Anti-HBs, D44: number analyzed (Participants) | 10 | 0
  Anti-HBs, D44 | 8447.1 [4040.7 to 17658.9] |
  Anti-HBs, D194: number analyzed (Participants) | 0 | 8
  Anti-HBs, D194 |  | 1996.3 [143.8 to 27707.6]

71. Secondary Outcome: Anti-Hepatitis B Surface (Anti-HBs) Antibody Concentrations in Serum - Step 2 Persistence
Description: as for outcome 70
Time Frame: At Day 0 (PRE) and post-vaccination (Day 44 for HBsAg/AS_2 Group and Day 194 for Engerix-B_2 Group)
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence (step 2 only) included all evaluable subjects, who complied with the protocol, for whom data concerning adaptive immunogenicity were available for at least one adaptive assay at Day 180 for the HBsAg/AS_2 Group and at Day 330 for the Engerix-B_2 Group.
Measure: Geometric Mean (95% Confidence Interval); unit: mIU/mL
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 10
mIU/mL
  Anti-HBs, PRE | 3.1 [3.1 to 3.1] | 3.1 [3.1 to 3.1]
  Anti-HBs, D44: number analyzed (Participants) | 10 | 0
  Anti-HBs, D44 | 8447.1 [4040.7 to 17658.9] |
  Anti-HBs, D194: number analyzed (Participants) | 0 | 10
  Anti-HBs, D194 |  | 2454.9 [311.4 to 19354.5]

72. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Step 2
Description: as for outcome 42
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each vaccine dose and across doses
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants
  Any Pain, Dose 1 | 10 | 3
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 3 | 0
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 2 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 10 | 10
  Any Pain, Dose 2 | 10 | 1
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Pain, Dose 2 | 2 | 0
  Any Redness, Dose 2: number analyzed (Participants) | 10 | 10
  Any Redness, Dose 2 | 2 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Redness, Dose 2 | 0 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 10 | 10
  Any Swelling, Dose 2 | 3 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 10
  Any Pain, Dose 3 |  | 1
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Pain, Dose 3 |  | 0
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 10
  Any Redness, Dose 3 |  | 0
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Redness, Dose 3 |  | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 10
  Any Swelling, Dose 3 |  | 0
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Swelling, Dose 3 |  | 0
  Any Pain, Across doses | 10 | 4
  Grade 3 Pain, Across doses | 2 | 0
  Any Redness, Across doses | 4 | 0
  Grade 3 Redness, Across doses | 0 | 0
  Any Swelling, Across doses | 3 | 0
  Grade 3 Swelling, Across doses | 0 | 0

73. Secondary Outcome: Number of Subjects With Any and Grade 3 Solicited Local Symptoms - Pooling Step
Description: as for outcome 42
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each vaccine dose and across doses
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 39
Participants
  Any Pain, Dose 1 | 28 | 10
  Grade 3 Pain, Dose 1 | 0 | 0
  Any Redness, Dose 1 | 9 | 1
  Grade 3 Redness, Dose 1 | 0 | 0
  Any Swelling, Dose 1 | 6 | 0
  Grade 3 Swelling, Dose 1 | 0 | 0
  Any Pain, Dose 2: number analyzed (Participants) | 37 | 38
  Any Pain, Dose 2 | 25 | 7
  Grade 3 Pain, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Pain, Dose 2 | 2 | 1
  Any Redness, Dose 2: number analyzed (Participants) | 37 | 38
  Any Redness, Dose 2 | 7 | 0
  Grade 3 Redness, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Redness, Dose 2 | 1 | 0
  Any Swelling, Dose 2: number analyzed (Participants) | 37 | 38
  Any Swelling, Dose 2 | 4 | 0
  Grade 3 Swelling, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Swelling, Dose 2 | 0 | 0
  Any Pain, Dose 3: number analyzed (Participants) | 0 | 10
  Any Pain, Dose 3 |  | 1
  Grade 3 Pain, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Pain, Dose 3 |  | 0
  Any Redness, Dose 3: number analyzed (Participants) | 0 | 10
  Any Redness, Dose 3 |  | 0
  Grade 3 Redness, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Redness, Dose 3 |  | 0
  Any Swelling, Dose 3: number analyzed (Participants) | 0 | 10
  Any Swelling, Dose 3 |  | 0
  Grade 3 Swelling, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Swelling, Dose 3 |  | 0
  Any Pain, Across doses | 31 | 12
  Grade 3 Pain, Across doses | 2 | 1
  Any Redness, Across doses | 12 | 1
  Grade 3 Redness, Across doses | 1 | 0
  Any Swelling, Across doses | 7 | 0
  Grade 3 Swelling, Across doses | 0 | 0

74. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms - Step 2
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise, myalgia, shivering and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination. At Day 0 of dose 2, two temperatures were collected: one at Hour 0 (H0) and a second one at Hour 18 (H18). The highest temperature between H0 et H18 was taken.
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each vaccine dose and across doses
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants
  Any Fatigue, Dose 1 | 8 | 3
  Grade 3 Fatigue, Dose 1 | 1 | 0
  Related Fatigue, Dose 1 | 7 | 2
  Any Gastrointestinal Symptoms, Dose 1 | 5 | 3
  Grade 3 Gastrointestinal Symptoms, Dose 1 | 1 | 0
  Related Gastrointestinal Symptoms, Dose 1 | 5 | 3
  Any Headache, Dose 1 | 7 | 4
  Grade 3 Headache, Dose 1 | 1 | 0
  Related Headache, Dose 1 | 7 | 3
  Any Malaise, Dose 1 | 5 | 0
  Grade 3 Malaise, Dose 1 | 1 | 0
  Related Malaise, Dose 1 | 5 | 0
  Any Myalgia, Dose 1 | 7 | 1
  Grade 3 Myalgia, Dose 1 | 0 | 0
  Related Myalgia, Dose 1 | 7 | 1
  Any Shivering, Dose 1 | 2 | 1
  Grade 3 Shivering, Dose 1 | 1 | 0
  Related Shivering, Dose 1 | 2 | 1
  Any Temperature, Dose 1 | 3 | 1
  Grade 3 Temperature, Dose 1 | 0 | 0
  Related Temperature, Dose 1 | 3 | 0
  Any Fatigue, Dose 2: number analyzed (Participants) | 10 | 10
  Any Fatigue, Dose 2 | 7 | 1
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Fatigue, Dose 2 | 1 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 10 | 10
  Related Fatigue, Dose 2 | 7 | 1
  Any Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 10 | 10
  Any Gastrointestinal Symptoms, Dose 2 | 3 | 0
  Grade 3 Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Gastrointestinal Symptoms, Dose 2 | 1 | 0
  Related Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 10 | 10
  Related Gastrointestinal Symptoms, Dose 2 | 3 | 0
  Any Headache, Dose 2: number analyzed (Participants) | 10 | 10
  Any Headache, Dose 2 | 6 | 0
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Headache, Dose 2 | 3 | 0
  Related Headache, Dose 2: number analyzed (Participants) | 10 | 10
  Related Headache, Dose 2 | 6 | 0
  Any Malaise, Dose 2: number analyzed (Participants) | 10 | 10
  Any Malaise, Dose 2 | 7 | 0
  Grade 3 Malaise, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Malaise, Dose 2 | 1 | 0
  Related Malaise, Dose 2: number analyzed (Participants) | 10 | 10
  Related Malaise, Dose 2 | 7 | 0
  Any Myalgia, Dose 2: number analyzed (Participants) | 10 | 10
  Any Myalgia, Dose 2 | 9 | 0
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Myalgia, Dose 2 | 0 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 10 | 10
  Related Myalgia, Dose 2 | 9 | 0
  Any Shivering, Dose 2: number analyzed (Participants) | 10 | 10
  Any Shivering, Dose 2 | 5 | 0
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 10 | 10
  Related Shivering, Dose 2 | 5 | 0
  Any Temperature, Dose 2: number analyzed (Participants) | 10 | 10
  Any Temperature, Dose 2 | 4 | 2
  Grade 3 Temperature, Dose 2: number analyzed (Participants) | 10 | 10
  Grade 3 Temperature, Dose 2 | 0 | 0
  Related Temperature, Dose 2: number analyzed (Participants) | 10 | 10
  Related Temperature, Dose 2 | 1 | 0
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Any Fatigue, Dose 3 |  | 1
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Fatigue, Dose 3 |  | 0
  Related Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Related Fatigue, Dose 3 |  | 1
  Any Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Any Gastrointestinal Symptoms, Dose 3 |  | 1
  Grade 3 Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Gastrointestinal Symptoms, Dose 3 |  | 0
  Related Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Related Gastrointestinal Symptoms, Dose 3 |  | 1
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Any Headache, Dose 3 |  | 2
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Headache, Dose 3 |  | 0
  Related Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Related Headache, Dose 3 |  | 2
  Any Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Any Malaise, Dose 3 |  | 0
  Grade 3 Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Malaise, Dose 3 |  | 0
  Related Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Related Malaise, Dose 3 |  | 0
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Any Myalgia, Dose 3 |  | 0
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Myalgia, Dose 3 |  | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Related Myalgia, Dose 3 |  | 0
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Any Shivering, Dose 3 |  | 0
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Shivering, Dose 3 |  | 0
  Related Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Related Shivering, Dose 3 |  | 0
  Any Temperature, Dose 3: number analyzed (Participants) | 0 | 10
  Any Temperature, Dose 3 |  | 0
  Grade 3 Temperature, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Temperature, Dose 3 |  | 0
  Related Temperature, Dose 3: number analyzed (Participants) | 0 | 10
  Related Temperature, Dose 3 |  | 0
  Any Fatigue, Across doses | 8 | 3
  Grade 3 Fatigue, Across doses | 2 | 0
  Related Fatigue, Across doses | 8 | 2
  Any Gastrointestinal Symptoms, Across doses | 6 | 4
  Grade 3 Gastrointestinal Symptoms, Across doses | 2 | 0
  Related Gastrointestinal Symptoms, Across doses | 6 | 4
  Any Headache, Across doses | 9 | 5
  Grade 3 Headache, Across doses | 4 | 0
  Related Headache, Across doses | 9 | 4
  Any Malaise, Across doses | 7 | 0
  Grade 3 Malaise, Across doses | 2 | 0
  Related Malaise, Across doses | 7 | 0
  Any Myalgia, Across doses | 9 | 1
  Grade 3 Myalgia, Across doses | 0 | 0
  Related Myalgia, Across doses | 9 | 1
  Any Shivering, Across doses | 6 | 1
  Grade 3 Shivering, Across doses | 1 | 0
  Related Shivering, Across doses | 6 | 1
  Any Temperature, Across doses | 6 | 3
  Grade 3 Temperature, Across doses | 0 | 0
  Related Temperature, Across doses | 3 | 0

75. Secondary Outcome: Number of Subjects With Any, Grade 3 and Related Solicited General Symptoms - Pooling Step
Description: Assessed solicited general symptoms were fatigue, gastrointestinal symptoms [nausea, vomiting, diarrhoea and/or abdominal pain], headache, malaise, myalgia, shivering and temperature [defined as oral temperature equal to or above (≥) 37.5 degrees Celsius (°C)]. Any = occurrence of the symptom regardless of intensity grade. Grade 3 symptom = symptom that prevented normal activity. Grade 3 fever = fever > 39.5 °C. Related = symptom assessed by the investigator as related to the vaccination. There was no pooling for temperature symptom between Step 1 and Step 2 due to difference in recording approach for the 18 hour data (nurse or self-assessment).
Time Frame: During the 7-day (Days 0-6) post-vaccination period following each vaccine dose and across doses
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 39
Participants
  Any Fatigue, Dose 1 | 11 | 9
  Grade 3 Fatigue, Dose 1 | 2 | 0
  Related Fatigue, Dose 1 | 9 | 8
  Any Gastrointestinal Symptoms, Dose 1 | 9 | 9
  Grade 3 Gastrointestinal Symptoms, Dose 1 | 1 | 1
  Related Gastrointestinal Symptoms, Dose 1 | 9 | 6
  Any Headache, Dose 1 | 21 | 9
  Grade 3 Headache, Dose 1 | 1 | 1
  Related Headache, Dose 1 | 18 | 7
  Any Malaise, Dose 1 | 9 | 2
  Grade 3 Malaise, Dose 1 | 1 | 0
  Related Malaise, Dose 1 | 9 | 2
  Any Myalgia, Dose 1 | 17 | 2
  Grade 3 Myalgia, Dose 1 | 0 | 0
  Related Myalgia, Dose 1 | 16 | 2
  Any Shivering, Dose 1 | 4 | 1
  Grade 3 Shivering, Dose 1 | 1 | 0
  Related Shivering, Dose 1 | 4 | 1
  Any Fatigue, Dose 2: number analyzed (Participants) | 37 | 38
  Any Fatigue, Dose 2 | 17 | 9
  Grade 3 Fatigue, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Fatigue, Dose 2 | 2 | 0
  Related Fatigue, Dose 2: number analyzed (Participants) | 37 | 38
  Related Fatigue, Dose 2 | 17 | 8
  Any Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 37 | 38
  Any Gastrointestinal Symptoms, Dose 2 | 7 | 5
  Grade 3 Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Gastrointestinal Symptoms, Dose 2 | 1 | 3
  Related Gastrointestinal Symptoms, Dose 2: number analyzed (Participants) | 37 | 38
  Related Gastrointestinal Symptoms, Dose 2 | 7 | 5
  Any Headache, Dose 2: number analyzed (Participants) | 37 | 38
  Any Headache, Dose 2 | 20 | 5
  Grade 3 Headache, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Headache, Dose 2 | 3 | 1
  Related Headache, Dose 2: number analyzed (Participants) | 37 | 38
  Related Headache, Dose 2 | 20 | 5
  Any Malaise, Dose 2: number analyzed (Participants) | 37 | 38
  Any Malaise, Dose 2 | 14 | 6
  Grade 3 Malaise, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Malaise, Dose 2 | 3 | 1
  Related Malaise, Dose 2: number analyzed (Participants) | 37 | 38
  Related Malaise, Dose 2 | 14 | 6
  Any Myalgia, Dose 2: number analyzed (Participants) | 37 | 38
  Any Myalgia, Dose 2 | 19 | 3
  Grade 3 Myalgia, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Myalgia, Dose 2 | 0 | 0
  Related Myalgia, Dose 2: number analyzed (Participants) | 37 | 38
  Related Myalgia, Dose 2 | 19 | 1
  Any Shivering, Dose 2: number analyzed (Participants) | 37 | 38
  Any Shivering, Dose 2 | 14 | 2
  Grade 3 Shivering, Dose 2: number analyzed (Participants) | 37 | 38
  Grade 3 Shivering, Dose 2 | 0 | 0
  Related Shivering, Dose 2: number analyzed (Participants) | 37 | 38
  Related Shivering, Dose 2 | 14 | 2
  Any Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Any Fatigue, Dose 3 |  | 1
  Grade 3 Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Fatigue, Dose 3 |  | 0
  Related Fatigue, Dose 3: number analyzed (Participants) | 0 | 10
  Related Fatigue, Dose 3 |  | 1
  Any Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Any Gastrointestinal Symptoms, Dose 3 |  | 1
  Grade 3 Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Gastrointestinal Symptoms, Dose 3 |  | 0
  Related Gastrointestinal Symptoms, Dose 3: number analyzed (Participants) | 0 | 10
  Related Gastrointestinal Symptoms, Dose 3 |  | 1
  Any Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Any Headache, Dose 3 |  | 2
  Grade 3 Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Headache, Dose 3 |  | 0
  Related Headache, Dose 3: number analyzed (Participants) | 0 | 10
  Related Headache, Dose 3 |  | 2
  Any Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Any Malaise, Dose 3 |  | 0
  Grade 3 Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Malaise, Dose 3 |  | 0
  Related Malaise, Dose 3: number analyzed (Participants) | 0 | 10
  Related Malaise, Dose 3 |  | 0
  Any Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Any Myalgia, Dose 3 |  | 0
  Grade 3 Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Myalgia, Dose 3 |  | 0
  Related Myalgia, Dose 3: number analyzed (Participants) | 0 | 10
  Related Myalgia, Dose 3 |  | 0
  Any Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Any Shivering, Dose 3 |  | 0
  Grade 3 Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Grade 3 Shivering, Dose 3 |  | 0
  Related Shivering, Dose 3: number analyzed (Participants) | 0 | 10
  Related Shivering, Dose 3 |  | 0
  Any Fatigue, Across doses | 18 | 12
  Grade 3 Fatigue, Across doses | 4 | 0
  Related Fatigue, Across doses | 18 | 11
  Any Gastrointestinal Symptoms, Across doses | 14 | 12
  Grade 3 Gastrointestinal Symptoms, Across doses | 2 | 4
  Related Gastrointestinal Symptoms, Across doses | 14 | 11
  Any Headache, Across doses | 26 | 11
  Grade 3 Headache, Across doses | 4 | 1
  Related Headache, Across doses | 24 | 10
  Any Malaise, Across doses | 15 | 7
  Grade 3 Malaise, Across doses | 4 | 1
  Related Malaise, Across doses | 15 | 7
  Any Myalgia, Across doses | 23 | 4
  Grade 3 Myalgia, Across doses | 0 | 0
  Related Myalgia, Across doses | 22 | 3
  Any Shivering, Across doses | 16 | 3
  Grade 3 Shivering, Across doses | 1 | 0
  Related Shivering, Across doses | 16 | 3

76. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Step 2
Description: as for outcome 45
Time Frame: Within the 28-day (Days 0-27) and post-vaccination period
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants | 5 | 4

77. Secondary Outcome: Number of Subjects With Any Unsolicited Adverse Events (AEs) - Pooling Step
Description: as for outcome 45
Time Frame: Within the 28-day (Days 0-27) post-vaccination period.
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 40
Participants | 20 | 19

78. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Step 2
Description: as for outcome 46
Time Frame: Up to Day 180 for the HBsAg/AS_2 Group and up to Day 330 for the Engerix-B_2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

79. Secondary Outcome: Number of Subjects With Serious Adverse Events (SAEs) - Pooling Step
Description: as for outcome 46
Time Frame: Up to Day 180 for the HBsAg/AS_1+2 Group and up to Day 330 for the Engerix-B_1+2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 40
Participants | 0 | 1

80. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Disorders (pIMDs) - Step 2
Description: as for outcome 47
Time Frame: Up to Day 180 for the HBsAg/AS_2 Group and up to Day 330 for the Engerix-B_2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants | 0 | 0

81. Secondary Outcome: Number of Subjects With Any Potential Immune-mediated Disorders (pIMDs) - Pooling Step
Description: as for outcome 47
Time Frame: Up to Day 180 for the HBsAg/AS_1+2 Group and up to Day 330 for the Engerix-B_1+2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 40
Participants | 0 | 0

82. Secondary Outcome: Number of Subjects With Any New Medical Conditions Requiring Medical Attention (MAEs) - Step 2
Description: MAEs were defined as events for which the subject received medical attention defined as hospitalization, an emergency room visit, or a visit to or from medical personnel (medical doctor) for any reason. Any MAE(s) = Occurrence of any MAE(s) regardless of intensity grade or relation to vaccination.
Time Frame: Up to Day 180 for the HBsAg/AS_2 Group and up to Day 330 for the Engerix-B_2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
Participants | 2 | 0

83. Secondary Outcome: Number of Subjects With Any New Medical Conditions Requiring Medical Attention (MAEs) - Pooling Step
Description: as for outcome 82
Time Frame: Up to Day 180 for the HBsAg/AS_1+2 Group and up to Day 330 for the Engerix-B_1+2 Group
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
Number analyzed (Participants) | 38 | 40
Participants | 2 | 1

84. Secondary Outcome: Levels of Alanine Aminotransferase (ALT) in Blood Samples - Step 2
Description: Biochemical laboratory parameters assessed included ALT levels. ALT concentrations were expressed in units per liter (U/L).
Time Frame: At Day 0 (PRE), Day 30, Day 32, Day 37, Day 60 for the HBsAg/AS_2 Group and Day 0 (PRE) Day 180, Day 182, Day 187 and Day 210 for the Engerix-B_2 Group
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
U/L
  ALT, PRE | 27.5 [23 to 33] | 31 [28 to 38]
  ALT, D30: number analyzed (Participants) | 10 | 0
  ALT, D30 | 25.5 [25 to 31] |
  ALT, D32: number analyzed (Participants) | 10 | 0
  ALT, D32 | 27 [20 to 36] |
  ALT, D37: number analyzed (Participants) | 10 | 0
  ALT, D37 | 23 [18 to 31] |
  ALT, D60: number analyzed (Participants) | 10 | 0
  ALT, D60 | 30 [23 to 33] |
  ALT, D180: number analyzed (Participants) | 0 | 10
  ALT, D180 |  | 34.5 [27 to 45]
  ALT, D182: number analyzed (Participants) | 0 | 9
  ALT, D182 |  | 31 [25 to 42]
  ALT, D187: number analyzed (Participants) | 0 | 9
  ALT, D187 |  | 34 [29 to 40]
  ALT, D210: number analyzed (Participants) | 0 | 10
  ALT, D210 |  | 29.5 [22 to 48]

85. Secondary Outcome: Levels of Aspartate Aminotransferase (AST) in Blood Samples - Step 2
Description: Biochemical laboratory parameters assessed included AST levels. AST concentrations were expressed in units per liter (U/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: U/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
U/L
  AST, PRE | 22.5 [21 to 24] | 28 [23 to 38]
  AST, D30: number analyzed (Participants) | 10 | 0
  AST, D30 | 22.5 [20 to 26] |
  AST, D32: number analyzed (Participants) | 10 | 0
  AST, D32 | 24 [22 to 26] |
  AST, D37: number analyzed (Participants) | 10 | 0
  AST, D37 | 20.5 [18 to 24] |
  AST, D60: number analyzed (Participants) | 10 | 0
  AST, D60 | 21.5 [18 to 31] |
  AST, D180: number analyzed (Participants) | 0 | 10
  AST, D180 |  | 25 [18 to 43]
  AST, D182: number analyzed (Participants) | 0 | 9
  AST, D182 |  | 29 [23 to 39]
  AST, D187: number analyzed (Participants) | 0 | 9
  AST, D187 |  | 25 [20 to 36]
  AST, D210: number analyzed (Participants) | 0 | 10
  AST, D210 |  | 22.5 [20 to 28]

86. Secondary Outcome: Levels of Basophils in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included basophil levels. Basophil levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Basophils, PRE | 0.04 [0.02 to 0.05] | 0.03 [0.02 to 0.04]
  Basophils, D30: number analyzed (Participants) | 10 | 0
  Basophils, D30 | 0.02 [0.01 to 0.07] |
  Basophils, D32: number analyzed (Participants) | 10 | 0
  Basophils, D32 | 0.04 [0.02 to 0.05] |
  Basophils, D37: number analyzed (Participants) | 10 | 0
  Basophils, D37 | 0.03 [0.01 to 0.06] |
  Basophils, D60: number analyzed (Participants) | 10 | 0
  Basophils, D60 | 0.05 [0.02 to 0.06] |
  Basophils, D180: number analyzed (Participants) | 0 | 10
  Basophils, D180 |  | 0.02 [0.01 to 0.04]
  Basophils, D182: number analyzed (Participants) | 0 | 9
  Basophils, D182 |  | 0.02 [0.01 to 0.04]
  Basophils, D187: number analyzed (Participants) | 0 | 9
  Basophils, D187 |  | 0.03 [0.02 to 0.05]
  Basophils, D210: number analyzed (Participants) | 0 | 10
  Basophils, D210 |  | 0.03 [0.01 to 0.04]

87. Secondary Outcome: Levels of Serum C Reactive Protein (CRP) in Blood Samples - Step 2
Description: Biochemical laboratory parameters assessed included CRP levels. CRP concentrations were expressed in milligrams per liter (mg/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
mg/L
  CRP, PRE | 5.55 [5 to 6.8] | 5.8 [5 to 9.5]
  CRP, D2 | 24.2 [16.6 to 32.7] | 5 [5 to 8.8]
  CRP, D30: number analyzed (Participants) | 10 | 0
  CRP, D30 | 6.8 [5.1 to 8.2] |
  CRP, D31: number analyzed (Participants) | 10 | 0
  CRP, D31 | 20.45 [10.4 to 21.9] |
  CRP, D32: number analyzed (Participants) | 10 | 0
  CRP, D32 | 33.75 [12.7 to 44.6] |
  CRP, D37: number analyzed (Participants) | 10 | 0
  CRP, D37 | 6.7 [5.5 to 10] |
  CRP, D60: number analyzed (Participants) | 10 | 0
  CRP, D60 | 5 [5 to 6.2] |
  CRP, D180: number analyzed (Participants) | 0 | 10
  CRP, D180 |  | 5.25 [5 to 6.8]
  CRP, D181: number analyzed (Participants) | 0 | 9
  CRP, D181 |  | 5 [5 to 6]
  CRP, D182: number analyzed (Participants) | 0 | 9
  CRP, D182 |  | 5 [5 to 7.3]
  CRP, D187: number analyzed (Participants) | 0 | 9
  CRP, D187 |  | 5 [5 to 6.7]
  CRP, D210: number analyzed (Participants) | 0 | 10
  CRP, D210 |  | 5 [5 to 7.8]

88. Secondary Outcome: Levels of Eosinophils in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included eosinophil levels. Eosinophil levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Eosinophils, PRE | 0.16 [0.09 to 0.23] | 0.18 [0.1 to 0.29]
  Eosinophils, D30: number analyzed (Participants) | 10 | 0
  Eosinophils, D30 | 0.17 [0.12 to 0.23] |
  Eosinophils, D32: number analyzed (Participants) | 10 | 0
  Eosinophils, D32 | 0.25 [0.17 to 0.33] |
  Eosinophils, D37: number analyzed (Participants) | 10 | 0
  Eosinophils, D37 | 0.19 [0.11 to 0.26] |
  Eosinophils, D60: number analyzed (Participants) | 10 | 0
  Eosinophils, D60 | 0.2 [0.09 to 0.26] |
  Eosinophils, D180: number analyzed (Participants) | 0 | 10
  Eosinophils, D180 |  | 0.14 [0.1 to 0.2]
  Eosinophils, D182: number analyzed (Participants) | 0 | 9
  Eosinophils, D182 |  | 0.17 [0.11 to 0.19]
  Eosinophils, D187: number analyzed (Participants) | 0 | 9
  Eosinophils, D187 |  | 0.18 [0.16 to 0.27]
  Eosinophils, D210: number analyzed (Participants) | 0 | 10
  Eosinophils, D210 |  | 0.16 [0.09 to 0.26]

89. Secondary Outcome: Levels of White Blood Cell (WBC) in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included white blood cells levels. WBC levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  WBC, PRE | 6.93 [5.51 to 9.67] | 5.67 [5.13 to 7.46]
  WBC, D30: number analyzed (Participants) | 10 | 0
  WBC, D30 | 6.41 [5.7 to 6.6] |
  WBC, D32: number analyzed (Participants) | 10 | 0
  WBC, D32 | 6.29 [5.24 to 8.09] |
  WBC, D37: number analyzed (Participants) | 10 | 0
  WBC, D37 | 6.37 [5.42 to 7.06] |
  WBC, D60: number analyzed (Participants) | 10 | 0
  WBC, D60 | 7.03 [5.65 to 8.5] |
  WBC, D180: number analyzed (Participants) | 0 | 10
  WBC, D180 |  | 6.02 [5.25 to 8.3]
  WBC, D182: number analyzed (Participants) | 0 | 9
  WBC, D182 |  | 6.15 [5.6 to 8.1]
  WBC, D187: number analyzed (Participants) | 0 | 9
  WBC, D187 |  | 7.35 [5.46 to 7.61]
  WBC, D210: number analyzed (Participants) | 0 | 10
  WBC, D210 |  | 5.91 [4.48 to 8.53]

90. Secondary Outcome: Levels of Lymphocytes in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included lymphocyte levels. Lymphocyte levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Lymphocytes, D0 | 2.13 [1.83 to 2.55] | 1.96 [1.69 to 2.37]
  Lymphocytes, D30: number analyzed (Participants) | 10 | 0
  Lymphocytes, D30 | 2.14 [1.8 to 2.47] |
  Lymphocytes, D32: number analyzed (Participants) | 10 | 0
  Lymphocytes, D32 | 1.7 [1.47 to 1.82] |
  Lymphocytes, D37: number analyzed (Participants) | 10 | 0
  Lymphocytes, D37 | 2.12 [1.98 to 2.32] |
  Lymphocytes, D60: number analyzed (Participants) | 10 | 0
  Lymphocytes, D60 | 2.12 [1.72 to 2.34] |
  Lymphocytes, D180: number analyzed (Participants) | 0 | 10
  Lymphocytes, D180 |  | 1.93 [1.84 to 2.45]
  Lymphocytes, D182: number analyzed (Participants) | 0 | 9
  Lymphocytes, D182 |  | 2.04 [1.75 to 2.44]
  Lymphocytes, D187: number analyzed (Participants) | 0 | 9
  Lymphocytes, D187 |  | 2.07 [1.76 to 2.27]
  Lymphocytes, D210: number analyzed (Participants) | 0 | 10
  Lymphocytes, D210 |  | 1.91 [1.46 to 2.94]

91. Secondary Outcome: Levels of Monocytes in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included monocyte levels. Monocyte levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Monocytes, D0 | 0.64 [0.47 to 0.74] | 0.5 [0.28 to 0.69]
  Monocytes, D30: number analyzed (Participants) | 10 | 0
  Monocytes, D30 | 0.54 [0.38 to 0.62] |
  Monocytes, D32: number analyzed (Participants) | 10 | 0
  Monocytes, D32 | 0.87 [0.8 to 1.07] |
  Monocytes, D37: number analyzed (Participants) | 10 | 0
  Monocytes, D37 | 0.47 [0.43 to 0.58] |
  Monocytes, D60: number analyzed (Participants) | 10 | 0
  Monocytes, D60 | 0.58 [0.49 to 0.68] |
  Monocytes, D180: number analyzed (Participants) | 0 | 10
  Monocytes, D180 |  | 0.46 [0.39 to 0.57]
  Monocytes, D182: number analyzed (Participants) | 0 | 9
  Monocytes, D182 |  | 0.43 [0.42 to 0.66]
  Monocytes, D187: number analyzed (Participants) | 0 | 9
  Monocytes, D187 |  | 0.44 [0.37 to 0.55]
  Monocytes, D210: number analyzed (Participants) | 0 | 10
  Monocytes, D210 |  | 0.52 [0.34 to 0.62]

92. Secondary Outcome: Levels of Neutrophils in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included neutrophil levels. Neutrophil levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Neutrophils, D0 | 4.02 [3.12 to 6.22] | 3.11 [2.3 to 4.56]
  Neutrophils, D30: number analyzed (Participants) | 10 | 0
  Neutrophils, D30 | 3.41 [2.87 to 3.93] |
  Neutrophils, D32: number analyzed (Participants) | 10 | 0
  Neutrophils, D32 | 3.42 [2.78 to 5.01] |
  Neutrophils, D37: number analyzed (Participants) | 10 | 0
  Neutrophils, D37 | 3.22 [2.76 to 3.9] |
  Neutrophils, D60: number analyzed (Participants) | 10 | 0
  Neutrophils, D60 | 4.18 [2.96 to 5.34] |
  Neutrophils, D180: number analyzed (Participants) | 0 | 10
  Neutrophils, D180 |  | 3.29 [2.99 to 4.67]
  Neutrophils, D182: number analyzed (Participants) | 0 | 9
  Neutrophils, D182 |  | 3.16 [2.89 to 4.88]
  Neutrophils, D187: number analyzed (Participants) | 0 | 9
  Neutrophils, D187 |  | 3.9 [3.18 to 4.29]
  Neutrophils, D210: number analyzed (Participants) | 0 | 10
  Neutrophils, D210 |  | 3.28 [2.29 to 4.88]

93. Secondary Outcome: Platelet Count in Blood Samples - Step 2
Description: Haematological laboratory parameters assessed included platelet count levels. Platelet count levels were expressed in billion cells per liter (billion cells/L).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: billion cells/L
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
billion cells/L
  Platelets, D0 | 269 [255 to 312] | 272 [215 to 322]
  Platelets, D30: number analyzed (Participants) | 10 | 0
  Platelets, D30 | 272.5 [215 to 330] |
  Platelets, D32: number analyzed (Participants) | 10 | 0
  Platelets, D32 | 257 [204 to 303] |
  Platelets, D37: number analyzed (Participants) | 10 | 0
  Platelets, D37 | 315.5 [286 to 330] |
  Platelets, D60: number analyzed (Participants) | 10 | 0
  Platelets, D60 | 282 [257 to 323] |
  Platelets, D180: number analyzed (Participants) | 0 | 10
  Platelets, D180 |  | 247 [237 to 276]
  Platelets, D182: number analyzed (Participants) | 0 | 9
  Platelets, D182 |  | 263 [248 to 274]
  Platelets, D187: number analyzed (Participants) | 0 | 9
  Platelets, D187 |  | 272 [260 to 280]
  Platelets, D210: number analyzed (Participants) | 0 | 10
  Platelets, D210 |  | 264.5 [214 to 314]

94. Secondary Outcome: Levels of Total Bilirubin in Blood Samples - Step 2
Description: Biochemical laboratory parameters assessed included total bilirubin levels. Bilirubin concentrations were expressed in milligrams per deciliter (mG/dL).
Time Frame: as for outcome 84
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
mg/dL
  Total Bilirubin, PRE | 0.4 [0.4 to 0.8] | 0.5 [0.3 to 0.7]
  Total Bilirubin, D2 | 0.45 [0.4 to 0.6] | 0.5 [0.3 to 1.5]
  Total Bilirubin, D30: number analyzed (Participants) | 10 | 0
  Total Bilirubin, D30 | 0.45 [0.3 to 0.8] |
  Total Bilirubin, D31: number analyzed (Participants) | 10 | 0
  Total Bilirubin, D31 | 0.55 [0.4 to 1] |
  Total Bilirubin, D32: number analyzed (Participants) | 10 | 0
  Total Bilirubin, D32 | 0.4 [0.2 to 0.6] |
  Total Bilirubin, D37: number analyzed (Participants) | 10 | 0
  Total Bilirubin, D37 | 0.45 [0.3 to 0.6] |
  Total Bilirubin, D60: number analyzed (Participants) | 10 | 0
  Total Bilirubin, D60 | 0.4 [0.3 to 0.6] |
  Total Bilirubin, D180: number analyzed (Participants) | 0 | 10
  Total Bilirubin, D180 |  | 0.45 [0.4 to 0.6]
  Total Bilirubin, D181: number analyzed (Participants) | 0 | 9
  Total Bilirubin, D181 |  | 0.6 [0.4 to 0.7]
  Total Bilirubin, D182: number analyzed (Participants) | 0 | 9
  Total Bilirubin, D182 |  | 0.6 [0.5 to 0.7]
  Total Bilirubin, D187: number analyzed (Participants) | 0 | 9
  Total Bilirubin, D187 |  | 0.5 [0.5 to 0.7]
  Total Bilirubin, D210: number analyzed (Participants) | 0 | 10
  Total Bilirubin, D210 |  | 0.6 [0.5 to 0.7]

95. Secondary Outcome: Levels of Diastolic Blood Pressure - Step 2
Description: Diastolic pressure was part of the list of vital signs followed at specific protocol-defined time points during this study, measured in millimeter of mercury (mmHg). On Days 30 and 180, diastolic blood pressure was assessed at multiple time points (plus 0 and 6 hours - H0, H6).
Time Frame: At Day 0 (PRE), Day 30 (H0, H6) at Day 31, at Day 32, at Day 37, at Day 60 for the HBsAg/AS_2 Group and at Day 0 (PRE), Day 180 (H0, H6), Day 181, at Day 182, at Day 187 and at Day 210 for the Engerix-B_2 Group
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
mmHg
  Diastolic, D0 | 74 [69 to 75] | 70 [67 to 72]
  Diastolic, D30 H0: number analyzed (Participants) | 10 | 0
  Diastolic, D30 H0 | 74.5 [73 to 78] |
  Diastolic, D30 H6: number analyzed (Participants) | 9 | 0
  Diastolic, D30 H6 | 71 [69 to 75] |
  Diastolic, D31: number analyzed (Participants) | 10 | 0
  Diastolic, D31 | 71.5 [68 to 78] |
  Diastolic, D32: number analyzed (Participants) | 10 | 0
  Diastolic, D32 | 71.5 [66 to 82] |
  Diastolic, D37: number analyzed (Participants) | 10 | 0
  Diastolic, D37 | 70 [69 to 76] |
  Diastolic, D60: number analyzed (Participants) | 10 | 0
  Diastolic, D60 | 72 [68 to 77] |
  Diastolic, D180 H0: number analyzed (Participants) | 0 | 10
  Diastolic, D180 H0 |  | 69 [63 to 71]
  Diastolic, D180 H6: number analyzed (Participants) | 0 | 10
  Diastolic, D180 H6 |  | 68.5 [65 to 71]
  Diastolic, D181: number analyzed (Participants) | 0 | 9
  Diastolic, D181 |  | 72 [66 to 75]
  Diastolic, D182: number analyzed (Participants) | 0 | 9
  Diastolic, D182 |  | 70 [69 to 72]
  Diastolic, D187: number analyzed (Participants) | 0 | 9
  Diastolic, D187 |  | 72 [64 to 77]
  Diastolic, D210: number analyzed (Participants) | 0 | 10
  Diastolic, D210 |  | 71.5 [65 to 74]

96. Secondary Outcome: Levels of Heart Rate - Step 2
Description: Heart rate was part of the list of vital signs followed at specific protocol-defined time points during this study. It was expressed in beats per minute. On Days 30 and 180, heart rate was assessed at multiple time points (plus 0 and 6 hours - H0, H6).
Time Frame: as for outcome 95
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: beats/minute
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
beats/minute
  Heart rate, PRE | 72 [63 to 80] | 70 [62 to 80]
  Heart rate, D30 H0: number analyzed (Participants) | 10 | 0
  Heart rate, D30 H0 | 70 [65 to 81] |
  Heart rate, D30 H6: number analyzed (Participants) | 9 | 0
  Heart rate, D30 H6 | 68 [64 to 77] |
  Heart rate, D31: number analyzed (Participants) | 10 | 0
  Heart rate, D31 | 84 [70 to 90] |
  Heart rate, D32: number analyzed (Participants) | 10 | 0
  Heart rate, D32 | 73 [67 to 83] |
  Heart rate, D37: number analyzed (Participants) | 10 | 0
  Heart rate, D37 | 65 [56 to 73] |
  Heart rate, D60: number analyzed (Participants) | 10 | 0
  Heart rate, D60 | 65 [62 to 72] |
  Heart rate, D180 H0: number analyzed (Participants) | 0 | 10
  Heart rate, D180 H0 |  | 71.5 [63 to 86]
  Heart rate, D180 H6: number analyzed (Participants) | 0 | 10
  Heart rate, D180 H6 |  | 70 [58 to 80]
  Heart rate, D181: number analyzed (Participants) | 0 | 9
  Heart rate, D181 |  | 81 [73 to 91]
  Heart rate, D182: number analyzed (Participants) | 0 | 9
  Heart rate, D182 |  | 72 [71 to 83]
  Heart rate, D187: number analyzed (Participants) | 0 | 9
  Heart rate, D187 |  | 78 [67 to 84]
  Heart rate, D210: number analyzed (Participants) | 0 | 10
  Heart rate, D210 |  | 76.5 [68 to 79]

97. Secondary Outcome: Levels of Respiratory Rate - Step 2
Description: Respiratory Rate was part of the list of vital signs followed at specific protocol-defined time points during this study. It was expressed as breaths per minute (breaths/min). On Days 30 and 180, respiratory rate was assessed at multiple time points (plus 0 and 6 hours - H0, H6).
Time Frame: as for outcome 95
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: breaths/min
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
breaths/min
  Respiratory rate, PRE | 12 [12 to 14] | 12 [12 to 14]
  Respiratory rate, D30 H0: number analyzed (Participants) | 10 | 0
  Respiratory rate, D30 H0 | 12.5 [11 to 13] |
  Respiratory rate, D30 H6: number analyzed (Participants) | 9 | 0
  Respiratory rate, D30 H6 | 12 [12 to 14] |
  Respiratory rate, D31: number analyzed (Participants) | 10 | 0
  Respiratory rate, D31 | 13 [12 to 14] |
  Respiratory rate, D32: number analyzed (Participants) | 10 | 0
  Respiratory rate, D32 | 12 [12 to 13] |
  Respiratory rate, D37: number analyzed (Participants) | 10 | 0
  Respiratory rate, D37 | 13.5 [12 to 14] |
  Respiratory rate, D60: number analyzed (Participants) | 10 | 0
  Respiratory rate, D60 | 12 [12 to 13] |
  Respiratory rate, D180 H0: number analyzed (Participants) | 0 | 10
  Respiratory rate, D180 H0 |  | 12.5 [12 to 15]
  Respiratory rate, D180 H6: number analyzed (Participants) | 0 | 10
  Respiratory rate, D180 H6 |  | 12.5 [12 to 14]
  Respiratory rate, D181: number analyzed (Participants) | 0 | 9
  Respiratory rate, D181 |  | 12 [12 to 14]
  Respiratory rate, D182: number analyzed (Participants) | 0 | 9
  Respiratory rate, D182 |  | 13 [12 to 14]
  Respiratory rate, D187: number analyzed (Participants) | 0 | 9
  Respiratory rate, D187 |  | 13 [12 to 15]
  Respiratory rate, D210: number analyzed (Participants) | 0 | 10
  Respiratory rate, D210 |  | 13.5 [12 to 15]

98. Secondary Outcome: Levels of Systolic Pressure - Step 2
Description: Systolic pressure was part of the list of vital signs followed at specific protocol-defined time points during this study, measured in millimeter of mercury (mmHg). On Days 30 and 180, systolic pressure was assessed at multiple time points (plus 0 and 6 hours - H0, H6).
Time Frame: as for outcome 95
Population: as for outcome 44
Measure: Median (Inter-Quartile Range); unit: mmHg
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 11
mmHg
  Systolic, PRE | 114 [110 to 116] | 112 [103 to 115]
  Systolic, D30 H0: number analyzed (Participants) | 10 | 0
  Systolic, D30 H0 | 114 [109 to 118] |
  Systolic, D30 H6: number analyzed (Participants) | 9 | 0
  Systolic, D30 H6 | 116 [104 to 121] |
  Systolic, D31: number analyzed (Participants) | 10 | 0
  Systolic, D31 | 112 [108 to 113] |
  Systolic, D32: number analyzed (Participants) | 10 | 0
  Systolic, D32 | 111.5 [102 to 116] |
  Systolic, D37: number analyzed (Participants) | 10 | 0
  Systolic, D37 | 108.5 [105 to 117] |
  Systolic, D60: number analyzed (Participants) | 10 | 0
  Systolic, D60 | 113 [104 to 122] |
  Systolic, D180 H0: number analyzed (Participants) | 0 | 10
  Systolic, D180 H0 |  | 111.5 [105 to 119]
  Systolic, D180 H6: number analyzed (Participants) | 0 | 10
  Systolic, D180 H6 |  | 111.5 [108 to 114]
  Systolic, D181: number analyzed (Participants) | 0 | 9
  Systolic, D181 |  | 115 [112 to 129]
  Systolic, D182: number analyzed (Participants) | 0 | 9
  Systolic, D182 |  | 117 [108 to 120]
  Systolic, D187: number analyzed (Participants) | 0 | 9
  Systolic, D187 |  | 112 [110 to 115]
  Systolic, D210: number analyzed (Participants) | 0 | 10
  Systolic, D210 |  | 112 [108 to 116]

99. Secondary Outcome: -Frequency of Hepatitis B Virus (HBs)-Specific Cluster of Differentiation (CD)4+ T-cells Expressing at Least 2 Immune Markers - Step 1
Description: Markers expressed were Interleukin-2 (IL-2), Interferon gamma (IFN-γ), Tumor Necrosis Factor (TNF)-α and Cluster of differentiation 40-Ligand (CD40L), as measured by classical (qualified assay) Intracellular Cytokine Staining (ICS),using frozen Peripheral blood mononuclear cells (PBMCs).
Time Frame: At Day 0 prior to vaccination (PRE) and Day 44 post-vaccination
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: T cells/million cells
Groups:
- Engerix-B_1 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30 followed by 3 doses of Engerix™- B vaccine at Day 0, Day 30 and Day 180. All vaccine were administered intramuscularly into the deltoid muscle of the non-dominant upper arm.
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 26 | 25
T cells/million cells
  PRE | 8 [1 to 52] | 1 [1 to 18]
  Day 44: number analyzed (Participants) | 26 | 24
  Day 44 | 4494 [2441 to 7494] | 268 [76 to 509]

100. Secondary Outcome: Frequency of Hepatitis B Virus (HBs)-Specific Cluster of Differentiation (CD)4+ T-cells Expressing at Least 2 Immune Markers - Step 1
Description: as for outcome 99
Time Frame: At Day 0 prior to vaccination (PRE), Day 44 and Day 180 post-vaccination
Population: The analysis was performed on the According-To-Protocol (ATP) cohort for persistence (step 1 only) included all evaluable subjects, who complied with the protocol, for whom data concerning adaptive immunogenicity were available for at least one adaptive assay at Day 180.
Measure: Median (Inter-Quartile Range); unit: T cells/ million cells
Groups:
- HBsAg/AS_1 Group: Subjects received, during Step 1 of the study, 1 dose of Placebo vaccine at Day -30, followed by 2 doses of HBsAg/AS vaccine, at Day 0 and Day 30. All vaccines were administered intramuscularly into the deltoid muscle of the nondominant upper arm.
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 24
T cells/ million cells
  PRE: number analyzed (Participants) | 26 | 24
  PRE | 8 [1 to 52] | 1 [1 to 21]
  Day 44: number analyzed (Participants) | 26 | 23
  Day 44 | 4494 [2441 to 7494] | 260 [33 to 527]
  Day 180: number analyzed (Participants) | 27 | 22
  Day 180 | 1119 [748 to 2181] | 34 [1 to 155]

101. Secondary Outcome: Frequency of Hepatitis B Virus (HBs)-Specific Cluster of Differentiation (CD)8+ T-cells Expressing at Least 2 Immune Markers - Step 1
Description: Markers expressed were Interleukin-2 (IL-2), Interferon gamma (IFN-γ), Tumor Necrosis Factor (TNF)-α and Cluste of differentiation 40-Ligand (CD40L), as measured by classical (qualified assay) Intracellular Cytokine Staining (ICS),using frozen Peripheral blood mononuclear cells (PBMCs).
Time Frame: At Day 0 prior to vaccination (PRE) and Day 44 post-vaccination
Population: as for outcome 41
Measure: Median (Inter-Quartile Range); unit: T cells/ million cells
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 26 | 25
T cells/ million cells
  PRE | 1 [1 to 24] | 1 [1 to 1]
  Day 44: number analyzed (Participants) | 26 | 24
  Day 44 | 38 [1 to 108] | 1 [1 to 33]

102. Secondary Outcome: Frequency of Hepatitis B Virus (HBs)-Specific Cluster of Differentiation (CD)8+ T-cells Expressing at Least 2 Immune Markers - Step 1
Description: as for outcome 99
Time Frame: At Day 0 prior to vaccination (PRE), Day 44 and Day 180 post-vaccination
Population: as for outcome 100
Measure: Median (Inter-Quartile Range); unit: T ceclls/ million cells
Arm/Group | HBsAg/AS_1 Group | Engerix-B_1 Group
Number analyzed (Participants) | 27 | 24
T ceclls/ million cells
  PRE: number analyzed (Participants) | 26 | 24
  PRE | 1 [1 to 24] | 1 [1 to 1]
  Day 44: number analyzed (Participants) | 26 | 23
  Day 44 | 38 [1 to 108] | 1 [1 to 42]
  Day 180: number analyzed (Participants) | 27 | 22
  Day 180 | 1 [1 to 17] | 1 [1 to 31]

103. Secondary Outcome: Number of Subjects With Solicited Symptoms, as Assessed by the Investigator/Study Nurse - Step 2
Description: as for outcome 44
Time Frame: Up to 3 days post-placebo/vaccine administration.
Population: as for outcome 44
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_2 Group | Engerix-B_2 Group
Number analyzed (Participants) | 10 | 10
Participants
  Pain, Dose 2: number analyzed (Participants) | 10 | 0
  Pain, Dose 2 | 8 | 0
  Pain, Dose 3: number analyzed (Participants) | 0 | 10
  Pain, Dose 3 | 0 | 1
  Redness, Dose 2: number analyzed (Participants) | 10 | 0
  Redness, Dose 2 | 5 | 0
  Redness, Dose 3: number analyzed (Participants) | 0 | 10
  Redness, Dose 3 | 0 | 0
  Swelling, Dose 2: number analyzed (Participants) | 10 | 0
  Swelling, Dose 2 | 3 | 0
  Swelling, Dose 3: number analyzed (Participants) | 0 | 10
  Swelling, Dose 3 | 0 | 0
  Induration, Dose 2: number analyzed (Participants) | 7 | 0
  Induration, Dose 2 | 1 | 0
  Induration, Dose 3: number analyzed (Participants) | 0 | 0
  Induration, Dose 3 | 0 | 0
  Fever, Dose 2: number analyzed (Participants) | 10 | 0
  Fever, Dose 2 | 0 | 0
  Fever, Dose 3: number analyzed (Participants) | 0 | 10
  Fever, Dose 3 | 0 | 0
  Muscle stiffness, Dose 2: number analyzed (Participants) | 10 | 0
  Muscle stiffness, Dose 2 | 7 | 0
  Muscle stiffness, Dose 3: number analyzed (Participants) | 0 | 10
  Muscle stiffness, Dose 3 | 0 | 1

104. Secondary Outcome: Number of Subjects With Solicited Symptoms, as Assessed by the Investigator/Study Nurse - Pooling Step
Description: as for outcome 44
Time Frame: Up to 3 days post-Dose 2 vaccine administration in HBsAg/AS_1+2 Group
Population: The analysis was performed on the Total Vaccinated cohort, of the HBsAg/AS_1+2 Group only, which included all subjects with the vaccine administration documented.
Measure: Count of Participants; unit: Participants
Arm/Group | HBsAg/AS_1+2 Group
Number analyzed (Participants) | 37
Participants
  Pain | 26
  Redness | 12
  Swelling | 7
  Induration: number analyzed (Participants) | 25
  Induration | 2
  Muscle stiffness | 22

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited symptoms: during the 28 Day (Days 0-27) post-vaccination period; SAEs: up to Day 180 for the HBsAg/AS_1+2 Group and up to Day 330 for the Engerix-B_1+2 Group.
Description: The safety analysis did not include subjects who received only the Placebo dose.
Arm/Group | HBsAg/AS_1+2 Group | Engerix-B_1+2 Group
All-Cause Mortality (participants affected / at risk) | 0/38 | 0/40
Serious Adverse Events (participants affected / at risk) | 0/38 | 1/40
Other Adverse Events (participants affected / at risk) | 16/38 | 13/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBsAg/AS_1+2 Group (N=38) | Engerix-B_1+2 Group (N=40)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | HBsAg/AS_1+2 Group (N=38) | Engerix-B_1+2 Group (N=40)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Dysmenorrhoea (Reproductive system and breast disorders) | 0 (0) | 3 (3)
Fatigue (General disorders) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 2 (3) | 5 (5)
Influenza like illness (General disorders) | 2 (2) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 1 (1)
Oral herpes (Infections and infestations) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.